# Portico<sup>™</sup> Re-sheathable Transcatheter Aortic Valve System US IDE Trial (PORTICO) NCT02000115

# Clinical Investigation Plan (CIP):

| Investigational Devices | |
|---|---|
| Description: | St. Jude Medical (SJM) Portico™ Transcatheter Aortic Valve |
| Trade Name: | Portico™ Transcatheter Heart Valve: |
| | Portico 23mm valve |
| | Portico 25mm valve |
| | Portico 27mm valve |
| | Portico 29mm valve |
| Model Numbers: | PRT-23-IDE or PRT-23 |
| | PRT-25-IDE or PRT-25 |
| | PRT-27-IDE |
| | PRT-29-IDE |
| | (or equivalent model numbers in respective geographies) |
| Associated Investigation Devices: | Portico Delivery Systems |
| | FlexNav Delivery Systems |
| | Portico Loading Systems |
| | FlexNav Loading Systems |
| Model Numbers: | PRT-DS-TF-18F-IDE, PRT-DS-TF-19F-IDE |
| | PRT-DS-ALT-18F-IDE, PRT-DS-ALT-19F-IDE |
| | PRT-LS-TFALT-18FID, PRT-LS-TFALT-19FID |
| | FN-DS-SM-IDE, FN-DS-LG-IDE, FN-LS-SM-IDE, FN-LS-LG- |
| | IDE(or equivalent model numbers in respective |
| | geographies) |
| Study Sponsor | |
| St. Jude Medical (now Abbott) | |
| National Co-Principal Investigators | National Co-Principal Investigators |
| <b>Document Version</b> | |
| Version: | |
| Date: | Date: August 8, 2018 |
| Version: | August 8, 2018 |

| Study Title: | Portico <sup>™</sup> Re-sheathable Transcatheter Aortic (PORTICO) | C Valve System US IDE Trial |
|---|---|---|
| CIP Number: | | |
| Study Device: | Portico™ Transcatheter Heart Valve and Deliv | very Systems |
| | ned, have read and understand the Clinical In ollow its content. | vestigation Plan specified above |
| Site Principal I | nvestigator Name (please print) | |
| Site Principal I | nvestigator Signature | <br>Date |

# **Table of Contents**

| 1 | PURPO | SE (PIVOTAL IDE AND CONTINUED ACCESS PROTOCOL (CAP)) | 7 |
|---|---|---|---|
| 1.: | 1 Indi | CATION FOR USE | 7 |
| 1.2 | 2 Stui | DY DESIGN AND OBJECTIVES | |
| | 1.2.1 | Study Design and Objectives (Pivotal IDE) | 7 |
| | 1.2.2 | Study Design and Objectives (CAP) | 8 |
| 1.3 | 3 Stui | PY ENDPOINTS (PIVOTAL IDE AND CAP) | 9 |
| | 1.3.1 | Pivotal IDE Endpoints (Randomized Cohort and Registries) | 9 |
| | 1.3.2 | Pivotal IDE FlexNav™ Study Endpoints | 10 |
| | 1.3.3 | CAP Endpoints | 11 |
| 1.4 | 4 SAM | PLE SIZE AND DURATION OF THE INVESTIGATION (PIVOTAL IDE AND CAP) | 11 |
| | 1.4.1 | Sample Size (Pivotal IDE) | |
| | 1.4.2 | Duration of the Investigation (Pivotal IDE) | 12 |
| | 1.4.3 | Sample Size (CAP) | |
| | 1.4.4 | Duration of the Investigation (CAP) | 12 |
| 2 | CLINIC | AL PROTOCOL (PIVOTAL IDE) | 12 |
| 2.: | 1 BAC | GROUND INFORMATION | |
| | 2.1.1 | Disease State and Patient Population | |
| | 2.1.2 | Therapy for Severe Aortic Stenosis | |
| | 2.1.3 | Transcatheter Aortic Valve Replacement | |
| | 2.1.4 | Status of TAVR in the United States | |
| | 2.1.5 | Valve-in-Valve | |
| | 2.1.6 | Updated Literature Search | |
| | 2.1.7 | Results of Literature Search | |
| | 2.1.8 | Primary Effectiveness Endpoint | |
| | 2.1.9 | Primary Safety Endpoint | |
| 2.2 | | MARY OF ST. JUDE MEDICAL PORTICO TRANSCATHETER VALVE CLINICAL EXPERIENCE | |
| 2.3 | 3 Rati | ONALE (PIVOTAL IDE AND CAP) | |
| | 2.3.1 | Pivotal IDE Rationale | 20 |
| | 2.3.2 | CAP Rationale | |
| 2.4 | 4 Nan | E AND DESCRIPTION OF THE INVESTIGATIONAL DEVICE (PIVOTAL IDE AND CAP) | 21 |
| 3 | PORTIC | O TRANSCATHETER AORTIC HEART VALVE | 22 |
| 3.3 | 1 Por | TICO DELIVERY SYSTEMS | |
| | 3.1.1 | First-Generation Portico Delivery System | |
| | 3.1.2 | Second-Generation FlexNav™ Delivery System | 24 |
| 3.2 | 2 Por | TICO INSTRUCTIONS FOR USE | 26 |
| 4 | RISK A | ND BENEFITS OF THE STUDY DEVICE AND CLINICAL STUDY (PIVOTAL IDE AND CAP) | 26 |
| 4.1 | | 5 | |
| 4.2 | | DER-BASED RISKS | |
| 4.3 | _ | MINIMIZATION | _ |
| 4.4 | 4 Beni | FITS | 30 |
| 5 | | POPULATION (PIVOTAL IDE AND CAP) | |
| 5.3 | | JSION CRITERIA | |
| 5.2 | | USION CRITERIA | |
| 5.3 | | ENING PROCESS | _ |
| | 5.3.1 | Additional Exclusion Criteria (Transcatheter Access-Related) | 35 |

| 6 | SL | JBJECT ASSIGNMENTS | 38 |
|---|---|---|---|
| | 6.1 | HIGH RISK COHORT (PIVOTAL IDE) | 38 |
| | 6.2 | EXTREME RISK COHORT (PIVOTAL IDE) | |
| | 6.3 | Valve-in-Valve Registry | |
| | 6.4 | Roll-in Registry | |
| | 6.5 | FLEXNAV STUDY | |
| | 6.6 | CONTINUED ACCESS PROTOCOL (CAP) | |
| | 6.7 | Screening | |
| | 6.8 | BASELINE ASSESSMENTS | 41 |
| | 6.9 | SUBJECT ENROLLMENT AND RANDOMIZATION | |
| 7 | ST | FUDY CONDUCT (PIVOTAL IDE AND CAP) | 44 |
| | 7.1 | Subject Informed Consent | |
| | 7.2 | SUBJECT SELECTION COMMITTEE | |
| | 7.2 | INDEX PROCEDURE | |
| | 7.4 | DISCHARGE VISIT (OR UP TO 7 DAYS POST PROCEDURE, WHICHEVER OCCURS FIRST) | |
| | 7.5 | FOLLOW-UP VISITS | |
| | 7.6 | 30 DAY VISIT (±7 DAYS) | |
| | 7.7 | 6 MONTH (±30 DAYS) (THIS VISIT IS NOT REQUIRED FOR CAP SUBJECTS ENROLLED UNDER VER. K OR LATER) | |
| | 7.8 | ONE-YEAR VISIT (-30 DAYS, + 45 DAYS) | |
| | 7.9 | ANNUAL VISITS (2 YEAR, 3 YEAR, 4 YEAR AND 5 YEAR (±60 DAYS)) | |
| | 7.10 | · | |
| | | 10.1 Unscheduled Visits for Evaluation of Suspected Neurological Event | |
| | 7.11 | EVALUATION OF ISCHEMIC STROKE AND MYOCARDIAL INFARCTION | |
| | 7.12 | SUBJECT WITHDRAWAL | |
| | 7.13 | TABLE OF ASSESSMENTS. | |
| | 7.14 | Study Activity Definitions | |
| | 7.15 | DETERMINATION OF THE AORTIC ANNULUS SIZE | |
| | 7.16 | CORE LABORATORIES | |
| | 7.17 | MEDICATIONS | |
| 8 | D | ATA COLLECTION AND MANAGEMENT (PIVOTAL IDE AND CAP) | |
| | 8.1 | SOURCE DATA AND SUBJECT FILES | |
| 9 | ΑI | DVERSE EVENTS (PIVOTAL IDE AND CAP) | 58 |
| | 9.1 | UNANTICIPATED ADVERSE DEVICE EFFECT | 58 |
| | 9.2 | ANTICIPATED ADVERSE EVENTS | 58 |
| | 9.3 | POTENTIAL ANTICIPATED ADVERSE EVENTS | 58 |
| | 9.4 | Adverse Event Reporting | 60 |
| | 9. | 4.1 Reporting All Adverse Events | 60 |
| | 9. | 4.2 Paravalvular Leak | |
| | 9. | 4.3 Reporting Unanticipated Adverse Device Effects | |
| | 9.5 | CLASSIFICATION OF CAUSAL RELATIONSHIPS | 61 |
| | 9.6 | SUBJECT DEATH | 61 |
| 10 | IN | IDEPENDENT BOARDS (PIVOTAL IDE AND CAP) | 61 |
| | 10.1 | CLINICAL EVENTS COMMITTEE | 61 |
| | 10.2 | DATA SAFETY MONITORING BOARD (DSMB) (PIVOTAL IDE) | 62 |
| 11 | ST | TATISTICAL METHODS AND ANALYSIS (PIVOTAL IDE) | 62 |
| | 11.1 | Analysis Populations | 62 |
| | 11.2 | RANDOMIZATION AND STRATIFICATION | 63 |

| | 44.3 | <b>D</b> | For a sure | 63 |
|---|---|---|---|---|
| | 11.3 | | ARY ENDPOINTS | |
| | 11.3 | | , ,, | |
| | <i>11.3</i><br>11.4 | | Primary Safety Endpoint LE SIZE CALCULATIONS | |
| | 11.4<br>11.4 | | Sample Size for the Primary Effectiveness Endpoint | |
| | 11.4. | _ | | |
| | | | Sample Size for the Primary Safety Endpoint Total Sample Size | |
| | <i>11.4.</i> .<br>11.5 | - | NDARY ENDPOINTS | |
| | 11.5<br>11.6 | | IPLICITY ADJUSTMENT | |
| | 11.0<br>11.7 | | TONAL ANALYSIS | |
| | 11.7<br>11.7. | | Subgroup Analysis: Sex/gender | |
| | 11.7 | | | |
| | 11.7 | | Additional Analyses of Primary Effectiveness Endpoint | |
| | 11.7. | | Additional Analyses of Primary Safety Endpoint | |
| | 11.7.4<br>11.8 | | ING ANALYSIS | |
| | | | TIONAL ASSESSMENT | |
| | 11.9<br>11.10 | | STICAL METHODS AND ANALYSIS (FLEXNAV STUDY, REGISTRIES AND CAP) | |
| 12 | STUD | Y TER | MINATION/WITHDRAWAL (PIVOTAL IDE AND CAP) | 73 |
| 13 | STLID | V N/A | NAGEMENT (PIVOTAL IDE AND CAP) | 75 |
| 13 | 3100 | | | |
| | 13.1 | | y Investigators | |
| | 13.2 | | DNAL PRINCIPAL INVESTIGATORS | |
| | 13.3 | | TIGATOR RESPONSIBILITIES | |
| | 13.4 | | RTS | |
| | 13.5 | | RDS | |
| | 13.6 | | rd Retention | |
| | 13.7 | | IDENTIALITY | |
| | 13.8 | | IDMENT PROCEDURE | |
| | 13.9 | | al Basis | |
| | 13.10 | | ANCE | _ |
| | 13.11 | | OPULATIONS | |
| | 13.12 | | RREPRESENTED GROUP CONSIDERATIONS | |
| | 13.13 | | y Monitoring | |
| | 13.14 | | LATORY INSPECTIONS | |
| | 13.15 | | PLIANCE | |
| | 13.16 | | OCOL DEVIATION | |
| | 13.17 | | E ACCOUNTABILITY | |
| | 13.18 | | OMIC AND QUALITY OF LIFE ANALYSIS | |
| | 13.19 | | CATIONS | |
| | 13.20 | | TIGATIONAL SITE START-UP | |
| | 13.20 | | Study Initiation Visit | |
| | 13.20 | ).2 | Site Activation | 86 |
| 14 | SPON | ISOR ( | CONTACT INFORMATION | 86 |
| 15 | BIBLI | UGRA | PHY | 87 |
| 16 | ADDE | NIDIC | rc | 01 |

# **List of Tables**

| TABLE 1. CLASSIFICATION OF SEVERITY OF AORTIC VALVE DISEASE IN ADULTS | 13 |
|---|---|
| Table 2. Mean Cumulative Rates of Effectiveness Endpoints | 16 |
| TABLE 3. MEAN CUMULATIVE RATES OF SAFETY ENDPOINTS ACROSS STUDIES | 16 |
| Table 4. Portico Transfemoral Valve Clinical Evaluation Series | 18 |
| TABLE 5. PRIMARY ENDPOINTS AND OBJECTIVES FOR PORTICO VALVE EVALUATIONS | 19 |
| TABLE 6. SUMMARY OF PORTICO TF VALVE EVALUATIONS AT 30 DAYS | 20 |
| TABLE 7. VALVE MODEL NUMBER AND REFERENCE DIMENSIONS | 21 |
| TABLE 8. DELIVERY AND LOADING SYSTEMS AND MODEL NUMBERS | 22 |
| TABLE 9. TABLE OF ASSESSMENTS (IDE PIVOTAL TRIAL AND CAP) | 50 |
| TABLE 10. STUDY ACTIVITY DEFINITIONS | |
| TABLE 11. SCHEDULE OF DATA COLLECTION (CASE REPORT FORMS) | |
| TABLE 12. REPORTING OBLIGATIONS. | |
| List of Figures | |
| FIGURE 1: PORTICO US PIVOTAL IDE TRIAL | |
| FIGURE 2. PORTICO TRANSCATHETER HEART VALVE | |
| FIGURE 3. FIRST-GENERATION PORTICO DELIVERY SYSTEM (DEPLOYMENT END) | |
| FIGURE 4. FIRST-GENERATION PORTICO DELIVERY SYSTEM | 24 |
| FIGURE 5: SECOND-GENERATION FLEXNAV™ DELIVERY SYSTEM HANDLE DETAIL | |
| FIGURE 6: SECOND- GENERATION FLEXNAV™ DELIVERY SYSTEM (PROXIMAL END) | 26 |
| FIGURE 7: STUDY CONDUCT FLOWCHART (PIVOTAL IDE AND CAP) | 37 |
| FIGURE 8. HIGH RISK COHORT FLOW CHART | 38 |
| FIGURE 9. EXTREME RISK COHORT FLOW CHART | 39 |
| FIGURE 10. PORTICO CLINICAL STUDY FLOW CHART | 43 |
| List of Appendices | |
| APPENDIX A: ABBREVIATIONS | |
| APPENDIX B: SYNOPSIS (PIVOTAL IDE) | |
| APPENDIX C: DEFINITIONS | |
| APPENDIX D: SURGICAL RISK ASSESSMENT TOOLS | |
| APPENDIX E: QUALITY OF LIFE – EQ-5D 3L | |
| APPENDIX F: QUALITY OF LIFE – SF-36v2 | |
| APPENDIX G: QUALITY OF LIFE – KANSAS CITY CARDIOMYOPATHY QUESTIONNAIRE (KCCQ) | |
| APPENDIX H: MINI-MENTAL STATE EXAMINATION (MMSE-2) | 115 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119<br>120 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119<br>120<br>122 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119<br>120<br>122<br>123 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 122 123 124 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 122 123 124 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 122 123 124 125 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 122 123 124 125 126 130 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 123 124 125 126 130 132 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 123 124 125 130 130 132 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 123 125 126 130 152 166 168 |
| APPENDIX I: CANADIAN CARDIOVASCULAR SOCIETY GRADING OF ANGINA PECTORIS | 119 120 123 125 126 130 152 166 168 |

#### 1 Purpose (Pivotal IDE and Continued Access Protocol (CAP))

#### 1.1 Indication for Use

The Portico™ Transcatheter Aortic Heart Valve is indicated for patients with symptomatic severe native aortic stenosis, who are considered high or extreme surgical risk.

#### 1.2 Study Design and Objectives

The PORTICO clinical study is an investigational device exemption (IDE) study comprised of the PORTICO pivotal IDE trial (pivotal IDE) and the PORTICO IDE Continued Access Protocol (CAP) study. The study design and objectives of these two separate study arms within the PORTICO clinical study are described below.

#### 1.2.1 Study Design and Objectives (Pivotal IDE)

The PORTICO pivotal IDE trial is a prospective, multi-center, randomized, controlled clinical investigation study designed to evaluate the safety and effectiveness of the SJM Portico Transcatheter Heart Valve and Delivery Systems (Portico) via transfemoral and alternative delivery methods in high-risk and extreme-risk patients.

As shown in Figure 1, the pivotal IDE trial includes a randomized cohort of 750 patients that will be used to support a Premarket Approval (PMA) application for the Portico™

Transcatheter Aortic Heart Valve in the United States. Prior to randomization, patients will be classified as high or extreme risk and stratified by vascular access within each risk group. At the time of the primary analysis, the risk cohorts will be combined.

There are two nested-registries within the pivotal IDE trial (Roll-in registry and Valve-in-Valve registry). Data from the IDE Valve-in-Valve registry will be used to support an expanded indication for transcatheter delivery of the Portico valve in a failed surgical bioprosthesis (TAVR-in-SAVR).

The objective of the FlexNav study

is to characterize the safety of the second-generation Portico Delivery System ("FlexNav™ Delivery System"). Thirty-day outcomes data from the FlexNav study will be used to support the PMA application for the Portico™ Transcatheter Aortic Heart Valve and the FlexNav™ Delivery System. A synopsis of the FlexNav study which includes details such as objectives, endpoints, and other study information is provided in Appendix W.

This protocol conforms to all the standards of Medicare coverage requirements. The PORTICO subject characteristics are consistent with Medicare population and the results are expected to be generalizable to the Medicare population.

Investigators enrolling subjects in the pivotal IDE trial under protocol version L or later will implant the Portico valve using the FlexNav™ Delivery System across all active study arms.



Figure 1: PORTICO US Pivotal IDE Trial

#### 1.2.2 Study Design and Objectives (CAP)

The PORTICO IDE Continued Access Protocol (CAP) study is a prospective, multicenter, single-arm investigational study designed to collect additional safety and clinical effectiveness data on the SJM Portico Transcatheter Aortic Heart Valve and Delivery System following completion of enrollment of subjects in the randomized cohort and FlexNav study of the PORTICO pivotal IDE trial.



Conduct of the CAP will follow the same protocol outlined for the pivotal IDE trial except where indicated. The main differences between the CAP and pivotal IDE trial include:

- A 6-month visit is not required for CAP subjects
- CAP subjects will not be randomized. All CAP subjects will receive a Portico device.
- The 6 Minute Walk Test (6MWT) and SF-36 questionnaire will not be required at any follow-up visit for CAP subjects.

A synopsis of the CAP which includes details such as objectives, endpoints, and other study information are provided in Appendix V.

#### 1.3 Study Endpoints (Pivotal IDE and CAP)

# 1.3.1 Pivotal IDE Endpoints (Randomized Cohort and Registries)

**Primary Effectiveness Endpoint:** A composite of all-cause mortality or disabling stroke at one year.

**Primary Safety Endpoint:** Non-hierarchical composite of all-cause mortality, disabling stroke, life threatening bleeding requiring blood transfusion, acute kidney injury requiring dialysis, or major vascular complications at 30 days.

# **Secondary Endpoints:**

- 1. Severe aortic regurgitation (AR) at one year
- 2. Kansas City Cardiomyopathy Questionnaire (KCCQ) at one year
- 3. Moderate or severe aortic regurgitation at one year
- 4. Six-minute walk at one year

#### **Descriptive Endpoints:**

- 1. Acute device success defined as:
  - Absence of procedural mortality AND
  - Correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  - Intended performance of the prosthetic heart valve (mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, no moderate or severe prosthetic valve regurgitation) AND
  - Successful access was obtained as intended by group assignment
- Kansas City Cardiomyopathy Questionnaire (KCCQ) at one year for Centers for Medicare and Medicaid Services (CMS) National Coverage Decision primary quality of life endpoint
- 3. Major vascular complications at 30 days from the index procedure
- 4. NYHA functional classification at 30 days, 6 months, and one year
- 5. Six-minute walk test at 30 days, 6 months, and one year
- 6. Paravalvular Leak (PVL) at 30 days, 6 months, and one year

- 7. Aortic insufficiency greater than trace at 30 days, 6 months, one year, and two years
- 8. Reintervention to treat aortic insufficiency at 1 year and 2 years
- 9. Permanent pacemaker insertion at 30 days from the index procedure
- 10. Major bleeding at 30 days from the index procedure
- 11. Acute kidney injury at 30 days from the index procedure
- 12. Individual components of the primary effectiveness endpoint
  - o All-cause mortality at 30 days, 6 months, one year and two years
  - o Disabling stroke at 30 days, 6 months, one year and two years
- 13. Non-disabling Stroke and Transient Ischemic Attack (TIA) at 30 days, 6 months, one year, and two years
- 14. Atrial fibrillation at one year and two years
- 15. Quality of Life (QOL) from baseline to 30 days, 6 months and one year

### 1.3.2 Pivotal IDE FlexNav™ Study Endpoints

**Primary Safety Endpoint:** VARC II defined major vascular complication rate at 30 days.

#### **Descriptive Endpoints:**

- Non-hierarchical composite of all-cause mortality, disabling stroke, life threatening bleeding requiring blood transfusion, acute kidney injury requiring dialysis, or major vascular complications at 30 days from the index procedure
- 2. All-cause mortality at 30 days and one year from the index procedure
- 3. Disabling stroke at 30 days and one year from the index procedure
- 4. Non-disabling stroke at 30 days from the index procedure
- 5. Life threatening bleeding requiring blood transfusion at 30 days from the index procedure
- 6. Major bleeding at 30 days from the index procedure
- 7. Acute kidney injury at 30 days from the index procedure
- 8. Minor vascular complication rates at 30 days from the index procedure
- 9. Permanent pacemaker insertion at 30 days from the index procedure
- 10. Paravalvular Leak (PVL) at 30 days from the index procedure
- 11. NYHA functional classification at 30 days from the index procedure
- 12. KCCQ Quality of Life (QoL) score from baseline to 30 days from the index procedure
- 13. Technical device success defined as successful vascular access, delivery and deployment of the Portico Valve; retrieval with the delivery system and correct positioning of a single valve in the proper anatomical location
- 14. Composite of all-cause mortality or disabling stroke at one year from the index procedure

#### 1.3.3 CAP Endpoints

**Primary Safety Endpoint:** A composite of VARC II defined all-cause mortality or disabling stroke at 30 days.

#### **Descriptive Endpoints:**

- Technical device success defined as successful vascular access, delivery and deployment of the Portico Valve; retrieval with the delivery system and correct positioning of a single valve in the proper anatomical location
- 2. Life threatening bleeding requiring blood transfusion and major bleeding at 30 days from the index procedure
- 3. Acute kidney injury at 30 days from the index procedure
- 4. Major and minor vascular access complication rate at 30 days from the index procedure
- 5. Permanent pacemaker insertion at 30 days from the index procedure
- 6. Paravalvular Leak (PVL) at 30 days and one year from the index procedure
- 7. NYHA functional classification at 30 days and one year from the index procedure
- 8. Disabling stroke at 30 days and one year from the index procedure
- 9. All-cause mortality at 30 days and one year from the index procedure
- 10. KCCQ Quality of Life (QOL) score from baseline to 30 days and one year from the index procedure





# 2 Clinical Protocol (Pivotal IDE)

# 2.1 Background Information

# 2.1.1 Disease State and Patient Population

Aortic stenosis (AS) is currently the most common valvular disease in the Western population¹ and its prevalence tends to increase with age, being present in 4.6% of adults ≥75 years.² Aortic stenosis (AS) can be primarily attributed to rheumatic disease and senile

degenerative calcification. Senile degenerative calcific AS is most common in the United States (U.S.) present in individuals older than 65 years. This calcification phenomenon is present in congenitally bicuspid or normal trileaflet valves. Calcific changes are due to an active disease process characterized by lipid accumulation, inflammation, and calcification.<sup>3,4</sup> This calcification process eventually leads to a restricted valve leaflet motion with obstruction to left ventricular outflow.<sup>3-5</sup>

Patients with AS are typically free from cardiovascular symptoms until late courses of the disease. However, once symptomatic, patients with severe AS have a poor prognosis, especially when combined with heart failure.<sup>5,7</sup>

Despite the tendency to grade the degree of AS based on a variety of hemodynamic measurements and natural history, ACC/AHA guideline authors describe aortic stenosis as a continuum.

The progression of AS can lead to the narrowing of aortic valve area by approximately 0.3 cm<sup>2</sup> per year. Also, the systolic pressure gradient across the valve can increase by as much as 15.19 mmHg per year. This functional deterioration of the aortic valve is more prevalent in the older population and usually coupled with coronary artery disease (CAD) and chronic renal insufficiency.<sup>8</sup>

Severe symptomatic AS is considered Class I indication for surgery. <sup>8,20</sup> The Joint ACC/AHA Task Force's published guidelines for the management of patients with valvular heart disease includes classification criteria for determining the severity of aortic stenosis (Table 1)<sup>20</sup>.

| Table 1. Classification of severity of aortic valve disease in adults | | | |
|---|---|---|---|
| Indicator | Mild | Moderate | Severe |
| Jet velocity (m/s) | < 3.0 | 3.0-4.0 | > 4.0 |
| Mean Gradient (mmHg) | < 25 | 25-40 | > 40 |
| Valve area (cm²) | > 1.5 | 1.0-1.5 | < 1.0 |
| Valve area index (cm²/m²) | | | < 0.6 |

After the onset of symptoms of angina pectoris, dyspnea, or syncope, annual mortality of patients with moderate-to-severe AS approaches 25%<sup>3</sup> and average survival is only 2 to 3 years. Other data also suggest the 2-year mortality rate can range from 44.4% for symptomatic AS patients<sup>9</sup> to as high as 79%<sup>10</sup> for predominant AS patients. Following symptomatic patients with severe aortic stenosis in whom operation was declined, O'Keefe<sup>11</sup> reported mortality rates of 45%, 63% and 75% at 1 year, 2 year, and 3 year follow-up, respectively. More recently, it has been established that inoperable patients with severe AS had a one year mortality rate of 50%.<sup>12</sup>

Relief of aortic valve obstruction typically results in an improvement of symptoms, hemodynamic parameters, and global left ventricle systolic function, as well as reversal of left ventricular hypertrophy.<sup>13</sup>

#### 2.1.2 Therapy for Severe Aortic Stenosis

Several treatment options are available to patients with symptomatic AS including optimal medical treatment. Until recently, surgical aortic valve replacement (SAVR) was the only effective treatment in adults with severe AS.<sup>8</sup> SAVR has been documented to significantly improve long-term survival in patients with AS.<sup>7,9,10</sup> Despite these proven positive outcomes of SAVR, the decision on whether to undergo SAVR can be influenced by prohibitive operative risk.<sup>9</sup>

Many patients with severe AS are considered high surgical risk and do not undergo SAVR due to severe comorbidities. Though some of these patients may be candidates for balloon valvuloplasty, this procedure has not offered any improvement in mortality. <sup>14</sup> SAVR has an average operative mortality of 3% to 8%, however primary patient characteristics and comorbidities, such as age and reduced left ventricular (LV) function, are associated with increased mortality within that range. <sup>15-18</sup> In addition, surgeon experience and hospital volume also affect outcomes with an absolute 2% lower mortality rate in the highest-volume compared with the lowest-volume hospitals. <sup>19</sup>

#### 2.1.3 Transcatheter Aortic Valve Replacement

A variety of conventional mechanical and bioprosthetic heart valves are readily accessible and commercially available in the U.S. However, some individuals are considered too high risk for open heart surgery, and may benefit from a less invasive procedure. With technological advancements, an alternative to SAVR, known as PAVR or TAVR (Percutaneous or Transcatheter Aortic Valve Replacement) and TAVI (Transcatheter Aortic Valve Implantation) has been under active investigation by a number of groups. <sup>21-28</sup> This concept was first demonstrated by Andersen et al<sup>29</sup> in 1992, who delivered a porcine bioprosthesis attached to a wire-based stent at various aortic sites with satisfactory hemodynamic results. In 2002, Cribier, et al, <sup>30</sup>reported the first successful human TAVR for the treatment of severe symptomatic aortic stenosis. Several single-center trials followed which demonstrated that this new approach was feasible for the treatment of severe aortic stenosis in patients who were inoperable or at a very high risk to undergo SAVR.

#### 2.1.4 Status of TAVR in the United States

The safety and effectiveness of TAVR has been confirmed with the recently published results of the Prospective, Randomized Placement of Aortic Transcatheter Valves (PARTNER) trial for high risk patients (Cohort A)<sup>34</sup> and inoperable patients (Cohort B)<sup>12</sup> (PMA # P100041). In 2011, with the FDA PMA approval of PARTNER Cohort A the Centers for Medicare and Medicaid Services (CMS) issued a coverage determination (NCD) for TAVR studies in the US (CAG-00430N).<sup>31</sup> The CMS national coverage decision provides requisite guidance on patient selection, post market surveillance methods and further clinical investigations of transcatheter aortic valve technologies in the extreme risk and high risk patient populations. The PARTNER trial has provided definitive data confirming TAVR as an alternative to SAVR. TAVR was found to be non-inferior to SAVR in both Cohort A (High Risk

patients) and Cohort B (Inoperable Risk patients) with severe aortic stenosis. When compared with standard therapy, TAVR significantly reduced the rates of all-cause mortality or repeat hospitalization, and cardiac symptoms, despite the higher incidence of major strokes and major vascular events, in the inoperable patients with severe AS.<sup>31</sup>

#### 2.1.5 Valve-in-Valve

There is a growing need for treatment options for patients with a failed bioprosthetic valve as the population ages, life expectancy improves, and the use of bioprosthetic valves increases. Operative mortality for elective redo aortic valve surgery is generally low (2% to 7%), but it can increase to more than 30% in high-risk and non-elective patients. Because transcatheter aortic valve (TAV)-in-surgical aortic valve (SAV) implantation represents a minimally invasive alternative to conventional redo surgery, it may prove to be as safe and effective as a redo surgery. Prospective comparisons with a large number of patients and long-term follow-up are required to confirm these potential advantages.

The most common reasons for an aortic valve implant redo, or valve-in-valve, are 1) wear and tear, 2) calcific degeneration, 3) pannus, 4) endocarditis, and 5) thrombus, where calcification and wear and tear are the most common reasons for bioprosthetic valve failure.<sup>36</sup>





# 2.1.8 Primary Effectiveness Endpoint



# 2.1.9 Primary Safety Endpoint




# 2.2 Summary of St. Jude Medical Portico Transcatheter Valve Clinical Experience









#### 2.3 Rationale (Pivotal IDE and CAP)

#### 2.3.1 Pivotal IDE Rationale

The rationale for this study is to potentially offer a SJM transcatheter Portico valve that is safe and effective for subjects with symptomatic, severe aortic valve stenosis who are considered at high or extreme risk for conventional surgical aortic valve replacement.

The rationale for conducting the FlexNav study as a separate arm of the pivotal IDE trial is to enable the direct comparison of 30-day safety outcomes data for the FlexNav™ Delivery System to the first-generation Portico Delivery System. Results from the FlexNav study will be included in a PMA application to support US approval of the Portico Transcatheter Heart Valve and FlexNav™ Delivery System.

#### 2.3.2 CAP Rationale

The rationale for the CAP is to allow current IDE study implanters to maintain their technical proficiency in Portico device implantation.

#### 2.4 Name and Description of the Investigational Device (Pivotal IDE and CAP)

The investigational devices used in the PORTICO clinical study consist of the Portico™ Transcatheter Aortic Heart Valve, the first-generation Portico Delivery System and the FlexNav™ Delivery System.

The PORTICO clinical study is utilizing the 23mm, 25mm, 27mm and the 29mm St. Jude Medical Portico™ Transcatheter Aortic Heart Valve. The Portico valve will be implanted using the Transfemoral access (TF), or alternative access (AA) consisting of Subclavian/Axillary and Transaortic access.

The Portico valve model number and reference dimensions are provided Table 7. Model numbers for equivalent devices may vary based on respective geographies.

| Table 7. Valve Model Number and Reference Dimensions | |
|---|---|
| Model Number | Intended to Treat Aortic Annulus Diameter |
| PRT-23-IDE | 19 – 21mm |
| PRT-25-IDE | 21 – 23mm |
| PRT-27-IDE | 23 – 25mm |
| PRT-29-IDE | 25 – 27mm |

The model numbers of the first-generation and second-generation ("FlexNav") Portico delivery systems and loading systems associated with the Portico valve are provided in Table 8. Part numbers are subject to change, but SJM maintains a list, which is available upon request. Model numbers for equivalent delivery and loading systems may vary based on respective geographies.

| Table 8. Delivery and Loading Systems and Model Numbers | |
|---|---|
| Model Number | Delivery System Diameter |
| PRT-DS-TF-18F-IDE | 18 Fr |
| PRT-DS-ALT-18F-IDE | 18 Fr |
| FN-DS-SM-IDE <sup>1</sup> | 18 Fr |
| PRT-DS-TF-19F-IDE | 19 Fr |
| PRT-DS-ALT-19F-IDE | 19 Fr |
| FN-DS-LG-IDE <sup>1</sup> | 19 Fr |
| PRT-LS-TFAL-18FID | N/A (loading system) |
| FN-LS-SM-IDE <sup>2</sup> | N/A (loading system) |
| PRT-LS-TFALT-19FID | N/A (loading system) |
| FN-LS-LG-IDE <sup>2</sup> | N/A (loading system) |
| ¹Indicates second-generation FlexNav™ Delivery System. Only allowed under protocol version L or later | |

<sup>2</sup>Indicates second-generation FlexNav™ Loading System. Only allowed under protocol version L or later

#### 3 Portico Transcatheter Aortic Heart Valve

The Portico Transcatheter Aortic Heart Valve (Figure 2) is designed to be implanted in the native aortic heart valve without open heart surgery and without concomitant surgical removal of the failed native valve.

The valve stent is made from nitinol, a material that has self-expanding properties and is radiopaque. The valve cuff is made from porcine pericardium that is sutured to the stent frame.

The cuff provides the sealing area for implantation. The valve orifice is made by suturing three valve leaflets, each made from a single layer of bovine pericardium, into a trileaflet configuration on the stent frame. The cuff and leaflet pericardial tissue is preserved and crosslinked in glutaraldehyde. Glutaraldehyde, formaldehyde and ethanol are used in the valve sterilization process.

The valve leaflets and valve cuff are processed using Linx™ anti-calcification treatment. The valve is supplied sterile and non-pyrogenic.



**Figure 2. Portico Transcatheter Heart Valve** 

# 3.1 Portico Delivery Systems

# 3.1.1 First-Generation Portico Delivery System

The first-generation Portico Delivery System is an over-the-wire, 0.035"-compatible system with an outer diameter ranging between 18 French (Fr) and 19 Fr depending on valve size.



Figure 3. First-Generation Portico Delivery System (deployment end)







Figure 4. First-Generation Portico Delivery System



The first-generation Portico Delivery System model number and reference dimensions are provided in the Instruction For Use (IFU) of the Portico™ Transcatheter Aortic Heart Valve.

# 3.1.2 Second-Generation FlexNav™ Delivery System

The second-generation FlexNav<sup>M</sup> Delivery System ("FlexNav Delivery System") is an overthe-wire, 0.035"- compatible system that includes a hydrophilic-coated, integrated sheath to facilitate gradual, controlled deployment of the valve in patients with a minimum vessel diameter of  $\geq$ 5mm.





Figure 5: Second-Generation FlexNav™ Delivery System Handle Detail







#### 3.2 Portico Instructions for Use

For instructions for use (IFU) of the Portico valve and the associated delivery and loading systems please refer to the following IFUs (Note: Model numbers for equivalent devices may vary based on respective geographies):

- Portico<sup>™</sup> Transcatheter Heart Valve (Models PRT-23-IDE, PRT-25-IDE, PRT-27-IDE, and PRT-29-IDE)
- Portico<sup>™</sup> Transfemoral Delivery Systems (Model PRT-DS-TF-18F-IDE and PRT-DS-TF-19F-IDE)
- Portico<sup>™</sup> Alternative Access Delivery Systems (Model PRT-DS-ALT-18F-IDE and PRT-DS-ALT-19F-IDE)
- Portico<sup>™</sup> Transfemoral/Alternative Access Loading Systems (Model PRT-LS-TFALT-18FID and PRT-LS-TFALT-19FID)
- FlexNav<sup>™</sup> Delivery System (FN-DS-SM-IDE, FN-DS-LG-IDE)
- FlexNav<sup>™</sup> Loading System (FN-LS-SM-IDE, FN-LS-LG-IDE)

#### 4 Risk and Benefits of the Study Device and Clinical Study (Pivotal IDE and CAP)

Participation in the pivotal IDE and CAP is expected to be associated with a similar risk and benefits profile to other commercially-available TAVR systems.

Please refer to the IFU of the Portico Transcatheter Aortic Heart Valve (which includes a description of risks and benefits), the risks listed below and to the adverse events section in this protocol for a list of the potential adverse events.

#### 4.1 Risks

There are potential risks associated with the use of transcatheter procedure with the study valve and commercially available control transcatheter valves. The potential risks include but are not limited to, the following:

- Access site complications (e.g., pain, bleeding, infection, hematoma, pseudoaneurysm, etc.)
- Acute coronary obstruction
- Acute myocardial infarction
- Access site injury
- Allergic reaction to antiplatelet agents, contrast medium, anesthesia, or valve components
- Anaphylactic shock/toxic reaction
- Annulus rupture
- Aortic rupture
- Ascending aorta trauma
- Atrio-ventricular node block
- AV fistula
- Bleeding
- Cardiac arrhythmias
- Cardiovascular or vascular injury, such as perforation or damage (dissection) of vessels, ventricle, myocardium or valvular structures that may require intervention
- Conduction system injury
- Death
- Endocarditis
- · Embolism: air, calcification or thrombus
- Exercise intolerance (weakness)
- Fever
- · Heart failure
- Hematoma
- Hemodynamic compromise
- Hemolysis
- Hemolytic anemia
- Hemorrhage
- Hypotension or hypertension
- Immunological reaction
- Infection
- Leakage, regurgitation
- Left ventricular failure/rupture

- Left ventricular impairment (due to apical scar)
- Myocardial ischemia
- Mitral valve insufficiency
- Multi-organ failure
- Neurological changes including stroke/transient ischemic attack;
- Non-structural dysfunction (i.e., entrapment by pannus, paravalvular leak, inappropriate sizing or positioning)
- Pannus
- Paravalvular leak
- Pericardial effusion
- Perforation of the myocardium or a blood vessel
- Potential coronary obstruction
- Renal failure
- Renal insufficiency
- Respiratory failure (shortness of breath)
- Sepsis
- Septal rupture
- Stenosis (high gradient)
- Stroke
- Structural valve deterioration (i.e., calcification, leaflet tear)
- Systemic peripheral ischemia
- Tamponade
- Valve explant
- Valve embolization
- Valve migration or malposition
- Valve stenosis
- Valve thrombosis
- Ventricular failure (acute)
- Ventricular rupture
- Vessel dissection or spasm

It is possible these complications could lead to:

- Transfusion
- Conversion to open surgical procedure
- Reoperation
- Emergent balloon valvuloplasty
- Emergent percutaneous coronary intervention (PCI)
- Emergent surgery (i.e., coronary artery bypass, heart valve replacement)
- Explantation
- Permanent disability
- Death
- Permanent pacemaker

All the listed risks may include the symptoms associated with the above mentioned medical conditions.

#### 4.2 Gender-Based Risks

A TAVR literature and background information search, pertaining to sex or gender differences in the intended patient population, did not reveal either a gender disparity favoring one gender over the other, or a race or ethnic disparity. This review shows that in over 50 studies, the median female percentage is 52% with a maximum of 94% female participation.<sup>39</sup> It is however evidenced in the literature that the risks experienced in TAVR can be observed in a higher rate within the female groups. The CoreValve ADVANCE<sup>40</sup> study revealed that females experienced a higher rate of stroke, major vascular complications, and major bleeding. Similarly, Buchanan et al. (2011) concluded that female sex was a predictor of major vascular complications with females requiring more transfusion. No differences were noted amongst patients undergoing TAVI in composite safety and efficacy endpoints according to sex.<sup>41</sup> Female subjects, however, had a better 1 year survival rate in the Sapien PARTNER trial.<sup>12,34</sup> Also, Humphries et al. (2012) in a study of 641 consecutive patients (51.3% female) showed that female gender is associated with better short- and long-term survival after TAVR. This is also evidenced in the PARTNER 1A findings.





#### 4.4 Benefits

There are no guaranteed benefits from participation in this study. Implantation of the transcatheter heart valve in the annular position may result in one or more of the following: improved valvular function, acute alleviation of symptoms related to aortic stenosis, improved morbidity and mortality.

Additionally, information gained from the conduct of this study may be of benefit to other people with the same medical condition in the future. The long-term results of using the study valve are not known at the present time. Alternative treatments include palliative medical therapy, aortic balloon valvuloplasty, transcatheter aortic valve delivery and surgical replacement of the aortic valve.

#### 5 Study Population (Pivotal IDE and CAP)

The PORTICO clinical study is limited to two subject cohorts with severe, symptomatic aortic stenosis who are determined to be at high or extreme operative risk for surgical aortic valve replacement. The operative risk determination of study candidates will be based on the Society of Thoracic Surgeons (STS) Adult Cardiac Surgery Risk Calculator. Subject case review

will be conducted by the Subject Selection Committee to determine the patient's eligibility to receive Portico valve.

These subject cohorts are defined as follows:

#### High risk cohort:

The **high risk** cohort is defined as subjects with severe aortic stenosis symptoms for whom conventional aortic valve replacement surgery is associated with high risk equivalent to an STS risk score that is  $\geq 8\%$ .

#### Extreme risk cohort:

The **extreme risk** cohort is defined as subjects with severe aortic stenosis symptoms and deemed unsuitable for conventional aortic valve replacement because of predicted probability of ≥50% mortality, or at risk for a serious irreversible complication by 30 days.

The surgical risk of study candidates will be determined by the heart team's interventional cardiologist(s) and cardiac surgeon(s) assessments taking into consideration the STS Adult Cardiac Surgery Risk Calculator.<sup>35</sup>

#### 5.1 Inclusion Criteria

#### **High Risk Cohort:**

All candidates for the High Risk Cohort of this study must meet **all** the following inclusion criteria:

- Subjects must have co-morbidities such that the surgeon and cardiologist Co-Investigators concur that the predicted risk of operative mortality is ≥15% or a minimum STS score of 8%. A candidate who does not meet the STS score criteria of ≥ 8% can be included in the study if a peer review by at least two surgeons concludes and documents that the patient's predicted risk of operative mortality is ≥15%. The surgeon's assessment of operative comorbidities not captured by the STS score must be documented in the study case report form as well as in the patient medical record.
- 2. Subject is 21 years of age or older at the time of consent.
- 3. Subject has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s or Doppler Velocity Index <0.25 and an initial aortic valve area (AVA) of  $\leq$  1.0 cm<sup>2</sup>

- (indexed EOA  $\leq$  0.6 cm<sup>2</sup>/m<sup>2</sup>). (Qualifying AVA baseline measurement must be within 60 days prior to informed consent).
- 4. Subject has symptomatic aortic stenosis as demonstrated by NYHA Functional Classification of II, III, or IV.
- 5. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
- 6. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.
- 7. Subject's aortic annulus is 19-27mm diameter as measured by CT conducted within 12 months prior to informed consent. Note: if CT is contraindicated and/or not possible to be obtained for certain subjects, a 3D echo and non-contrast CT of chest and abdomen/pelvis may be accepted if approved by the subject selection committee.

#### **Extreme Risk Cohort:**

All candidates for the Extreme Risk Cohort of this study must meet # 2, 3, 4, 5, 6, 7 of the above criteria, *and* 

1. The subject, after formal consults by a cardiologist and two cardiovascular surgeons agree that medical factors preclude operation, based on a conclusion that the probability of death or serious, irreversible morbidity exceeds the probability of meaningful improvement. Specifically, the probability of death or serious, irreversible morbidity should exceed 50%. The surgeons' consult notes shall specify the medical or anatomic factors leading to that conclusion and include a printout of the calculation of the STS score to additionally identify the risks in these patients.

#### **All Candidates:**

Additionally, all candidates for the study must meet the following inclusion criteria for the TAVR Leaflet Motion Sub-study, until the minimum sub-study sample size has been achieved, as described in Appendix S. This sub-study is not applicable for subjects enrolled under protocol Version K or later (including CAP subjects) as the minimum sub-study sample size has been achieved:

Be willing and able to undergo, at both 30 days and 6 months post-implant, a Multi-Slice Computed Tomography (MSCT) scan (or TEE, if medically or technically contraindicated for a MSCT) of the heart and cardiac structures.

#### 5.2 Exclusion Criteria

#### **High and Extreme Risk Cohort:**

Candidates will be excluded from the study if **any** of the following conditions are present:

- 1. Evidence of an acute myocardial infarction (defined as: ST Segment Elevation as evidenced on 12 Lead ECG) within 30 days prior to index procedure.
- 2. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified as verified by echocardiography.
- 3. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation 3-4+).
- 4. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to index procedure.
- 5. Pre-existing prosthetic heart valve or other implant in any valve position, prosthetic ring, severe circumferential mitral annular calcification (MAC) which is continuous with calcium in the LVOT, severe (greater than 3+) mitral insufficiency, or severe mitral stenosis with pulmonary compromise. Subjects with pre-existing surgical bioprosthetic aortic heart valve should be considered for the Valve-in-Valve registry.
- 6. Blood dyscrasias as defined: leukopenia (WBC<3000 mm³), acute anemia (Hb < 9 g/dL), thrombocytopenia (platelet count <50,000 cells/mm³).
- 7. History of bleeding diathesis or coagulopathy.
- 8. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
- Untreated clinically significant coronary artery disease requiring revascularization.
- 10. Hemodynamic instability requiring inotropic support or mechanical heart assistance.
- 11. Need for emergency surgery for any reason.
- 12. Hypertrophic cardiomyopathy with or without obstruction (HOCM).
- 13. Severe ventricular dysfunction with LVEF <20% as measured by resting echocardiogram.
- 14. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
- 15. Active peptic ulcer or upper GI bleeding within 3 months prior to index procedure.
- 16. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine (Ticlid), or clopidogrel (Plavix), or sensitivity to contrast media which cannot be adequately premedicated.
- 17. Recent (within 6 months prior to index procedure date) cerebrovascular accident (CVA) or a transient ischemic attack (TIA).

- 18. Renal insufficiency (creatinine > 3.0 mg/dL) and/or end stage renal disease requiring chronic dialysis.
- 19. Life expectancy < 12 months from the time of informed consent due to non-cardiac co-morbid conditions.
- 20. Significant aortic disease, including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5cm or greater; marked tortuosity (hyperacute bend), aortic arch atheroma (especially if thick [> 5 mm], protruding or ulcerated) or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta (applicable for transfemoral patients only).
- 21. Native aortic annulus size < 19 mm or > 27 mm per the baseline diagnostic imaging.
- 22. Aortic root angulation > 70° (applicable for transfemoral patients only).
- 23. Currently participating in an investigational drug or device study.
- 24. Active bacterial endocarditis within 6 months prior to the index procedure.
- 25. Bulky calcified aortic valve leaflets in close proximity to coronary ostia.
- 26. Non-calcified aortic annulus
- 27. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath such as severe obstructive calcification, or severe tortuosity (applicable for transfemoral patients only).

#### **5.3** Screening Process

At the time the patient agrees to participate after receiving information and all the patient's questions have been answered satisfactorily, the study informed consent form will be signed. Patients who sign an informed consent form and meet all the inclusion criteria and none of the exclusion criteria will be reviewed and confirmed by the Subject Selection Committee for participation eligibility. Subject selection should take place within 30 days from the date the subject provided informed consent. Once the subject is selected to participate in the study, baseline assessments and randomization (if applicable) can be completed. The index procedure should take place no later than 14 calendar days from subject enrollment.

Subjects who meet the subject selection criteria and are confirmed by the Subject Selection Committee will be assigned to cohorts based on their surgical risk level and either randomized into the pivotal IDE randomized cohort or enrolled into a study-defined registry (Roll-in or Valve-in-Valve), the FlexNav study or the CAP. Subjects who do not meet the selection criteria will not be scheduled for an implant procedure and will not be considered enrolled into the study.

If a subject is consented and undergoes study-specific testing (i.e., testing that would not be done if they were not being considered for the study) but is not enrolled in the study, the

subject should be followed for adverse events for 30 days from informed consent and then withdrawn from study participation.

For subjects consented under protocol version L or later, if a subject undergoes study-specific testing but does not undergo a Portico implant attempt with the FlexNav™ Delivery System the subject will not be considered enrolled in the study and will not require any further follow-up.

Figure 7 summarizes subjects' screening and enrollment flow.

Subject screening depends on the joint collaboration of investigators (including designated interventional cardiologist(s) and designated cardiac surgeon(s)) at each site. All suitable subjects must undergo the established institutional specific multidisciplinary team assessment to confirm both appropriateness for transcatheter aortic valve placement and high-risk designation. Both a cardiologist investigator and a cardiac surgeon investigator must be involved in the subject selection and screening process. All subjects evaluated for severe aortic stenosis in medical and surgical departments that are high or extreme risk candidates for AVR should be screened for study eligibility.

The investigators are responsible for ensuring subject eligibility. Study sites will maintain a log of all the screened subjects and subjects enrolled. Reasons for meeting study criteria but failing to be enrolled will be captured on the screening log and may be monitored by SJM.

#### 5.3.1 Additional Exclusion Criteria (Transcatheter Access-Related)

For subjects who do not qualify for transfemoral access, the following exclusion criteria will be used to screen for an appropriate alternative access delivery method.

#### 5.3.1.1 Transaortic Subject Cohort Specific Exclusion Criteria

- 1. Subject has pre-existing patent RIMA graft that would preclude access.
- 2. Subject has a hostile chest or other condition that complicates transaortic access.
- 3. Subject has a porcelain aorta, defined as an extensive circumferential calcification of the ascending aorta that would complicate TAo access.

For subjects enrolled under version L of the protocol, the following exclusion criteria apply for transaortic access using the FlexNav™ Delivery System:

- Subject has a distance between the annular plane and the aortic access site <7 cm (2.8")
- 2. Subject has a distance between the annular plane and the separate introducer sheath distal tip <6 cm (2.4")

#### 5.3.1.2 Subclavian/Axillary Subject Cohort Specific Exclusion Criteria

- 1. Subject's access vessel (subclavian/axillary) diameter will not allow for introduction of the applicable 18 Fr or 19 Fr delivery system.
- 2. Subject's subclavian/axillary arteries have severe calcification and/or tortuosity.

- 3. Subject's aortic root angulation is:
  - Left Subclavian/Left Axillary: >70°
  - Right Subclavian/Right Axillary: >30°
- 4. Subject has a history of patent LIMA/RIMA graft that would preclude access

For subjects enrolled under version L of the protocol, the following exclusion criteria apply for subclavian/axillary access using the FlexNav™ Delivery System:

- 1. Subject's access vessel (subclavian/axillary) has a distance between the annular plane and the integrated sheath distal tip <17 cm (6.7")
- 2. Subject's access vessel requires the delivery system to be advanced through a separate introducer sheath

For selection of the appropriate alternative access method, subjects will be screened using the access specific exclusion criteria, and the selection of the alternative access method will be based on the evaluation by the site and the Subject Selection Committee.


Figure 7: Study Conduct Flowchart (Pivotal IDE and CAP)

# 6 Subject Assignments

Subjects will be assigned to one of the following cohorts:

# 6.1 High Risk Cohort (Pivotal IDE)

High risk subjects with an annular size between 19-27mm who qualify for transfemoral access and have a suitable iliofemoral vasculature for both Portico valve and an FDA approved commercially available transcatheter valve (CAV) will be randomized into the transfemoral arm to receive either the Portico valve or the CAV. Subjects who do not qualify for the transfemoral access arm (iliofemoral vasculature is not suitable for both Portico and CAV) will be randomized within the alternative access arm to receive either the Portico valve or CAV (Figure 8).



TF=Transfemoral, CAV= Commercially Available Transcatheter Valve, AA=Alternative Access

Figure 8. High Risk Cohort Flow Chart

# 6.2 Extreme Risk Cohort (Pivotal IDE)

Extreme risk subjects will be assigned to the Extreme Risk Cohort as follows:

Extreme risk subjects with annular size between 19-27mm who qualify for transfemoral access and have suitable iliofemoral vasculature suitable for both Portico and CAV will be randomized into the transfemoral arm to receive either the Portico valve or CAV. Subjects who do not qualify for the transfemoral access arm (iliofemoral vasculature is not suitable for both Portico and CAV) will be randomized within the alternative access arm to receive either the Portico valve or CAV (Figure 9).



TF=Transfemoral, CAV= Commercially Available Transcatheter Valve, AA=Alternative Access

**Figure 9. Extreme Risk Cohort Flow Chart** 

# 6.3 Valve-in-Valve Registry

Subjects who have documented failed aortic surgical valve prosthesis and are deemed eligible to receive a transcatheter Portico valve into the existing bioprosthesis will be considered for eligibility in the Valve-in-Valve registry. The Valve-in-Valve registry will enroll up to 100 qualified subjects from the pivotal IDE trial or CAP.

Valve-in-valve registry subjects must meet all the applicable inclusion criteria and none of the applicable exclusion criteria for the high or extreme risk cohort (Sections 5.1 & 5.2).

Examples of criteria that may not apply include inclusion criterion numbers **3** and **4** (the bioprosthetic valve may be stenotic or require replacement due to other forms of structural valve deterioration), and exclusion criterion numbers **2**, **3**, **5** (existing surgical bioprosthetic aortic valve), **21**, and **26**. If the subject has a bioprosthetic valve in another location, the subjects will be excluded from the PORTICO clinical study.

Valve-in-valve subjects' data will not be included in the randomized population nor the primary data analysis; however, the data will be analyzed and presented separately to support an expanded indication for Valve-in-Valve use (Portico-in-SAVR).

All Valve-in-Valve subjects enrolled under protocol version L or later will have a Portico valve implanted using the FlexNav<sup>™</sup> Delivery System. Implanting physicians will be required to have completed a minimum of one (1) roll-in subject in the FlexNav study before enrolling a subject in the IDE Valve-in-Valve registry.

# 6.4 Roll-in Registry

Prior to enrolling subjects in the pivotal IDE randomized cohort, sites will be required to complete a minimum of two (2) and up to three (3) roll-in patients per primary implanting physician. However, implanting physicians with prior Portico experience and with a minimum of 3 implants in the last 6 months will not be required to include roll-in patients.

For subjects enrolled under protocol version L or later, all primary implanting physicians irrespective of prior Portico implant experience will be required to complete a minimum of one (1) and up to three (3) roll-in patients using the FlexNav™ Delivery System.

All roll-in subjects will be added to the IDE Roll-in Registry. The roll-in subjects must meet all the inclusion criteria and none of the exclusion criteria and be approved by the Subject Selection Committee. These subjects will be followed per protocol for the duration of the study, or until subject's withdrawal or death. The roll-in subjects' data will not be included in the randomized population nor the primary data analysis; however, the data will be analyzed and presented separately.

# 6.5 FlexNav Study

High and extreme risk subjects with an annular size between 19-27mm with suitable anatomy for transfemoral or alternative access valve implantation using the FlexNav<sup>TM</sup> Delivery System (minimum vessel requirement  $\geq$  5mm) will be enrolled in the FlexNav study. All FlexNav study subjects will receive a Portico device (no randomization).

The number of roll-in patients required by a site before they can contribute to the FlexNav study will be at the discretion of the Sponsor. All roll-in subjects will be designated as such prior to enrollment and will be added to the IDE Roll-in Registry.

Following the successful completion of roll-in subjects, sites will enroll subjects into the FlexNav study. These enrolled subjects will be considered part of the 'analysis population'.

Analysis subject data (excluding roll-ins) will be summarized and presented separately to the randomized cohort in the PMA application.

#### 6.6 Continued Access Protocol (CAP)

After the pivotal IDE trial has met its minimum sample-size for the randomized cohort and the FlexNav study, sites may choose to participate in the CAP and enroll high and extreme risk subjects with an annular size between 19-27mm with suitable anatomy for transfemoral or alternative access valve implantation. All CAP subjects will receive a Portico valve (no randomization).

#### 6.7 Screening

Data available in the patient's medical record may be utilized to fulfill screening and baseline requirements and testing does not need to be repeated if performed within 60 days prior to informed consent. Computed Tomography (CT) scan with angiography and coronary and aortic angiogram (with runoff if clinically indicated) may be performed within 12 months prior to informed consent.

After subject informed consent is obtained, study-specific screening evaluation may be conducted to determine inclusion in the study. All cardiac medications and all medications given for cardiovascular effect may be continued at their prescribed dosages.

- 1. Demographics
- 2. Medical History
- 3. Canadian Cardiovascular Society (CCS) Angina Scale Assessment
- 4. Surgical Risk Assessment tools (STS Risk Score, and EuroSCORE II)
- 5. Forced Expiratory Volume (FEV1), if clinically indicated
- 6. Physical Exam
- 7. Echocardiography to include comprehensive transthoracic or transesophageal 2D echocardiogram, including assessment of aortic valve gradients (mean and peak), areas, indices, degree of regurgitation, cardiac output and cardiac index, left ventricle systolic function (global and segmental)
- 8. Lab Measurements (per Table 9, Table of Assessments)
- 9. 12 Lead Electrocardiogram (ECG)
- 10. Computed Tomography Scan with Angiography for chest, abdomen and pelvis: aortic root and valve annulus sizing, assessment of suitability of iliofemoral access, and determination of appropriate coaxial angles for optimizing the valve implantation procedure. CT scan performed up to 12 months prior to consent will be acceptable.
- 11. 3D Transesophageal Echocardiogram (TEE) if CT is contraindicated
- 12. New York Heart Association (NYHA) Functional Classification
- 13. Frailty Index Assessment
  - a. Katz Index of Activities of Daily Living
  - b. Grip strength
  - c. 15 ft. walk
- 14. Coronary and aortic angiogram (arteriograms of the lower abdominal aorta to the femoral arteries), with runoff if clinically indicated. Coronary and aortic angio performed up to 12 months prior to consent will be acceptable.

#### 6.8 Baseline Assessments

The following baseline data will be collected for all subjects prior to the index procedure.

- 1. Chest X-ray
- 2. Cardiovascular medications documentation
- 3. Modified Rankin Scale (mRS)
- 4. NIH Stroke Scale (NIHSS)
- 5. Barthel Index
- 6. Quality of Life Measures (QoL) (For CAP subjects enrolled under Ver. K or later, only the KCCQ and EQ-5D are required.)
- 7. MMSE-2:SV
- 8. Six Minute Walk Test (6MWT) (Not required for CAP subjects enrolled under Ver. K or later)

9. Troponin or CK/CK-MB, INR (if subject is on Coumadin or Warfarin)

# 6.9 Subject Enrollment and Randomization

All subjects who meet the study eligibility requirements will be assigned into an applicable registry (Roll-in or Valve-in-Valve), the FlexNav study, the CAP or one of the pivotal IDE randomized cohorts for operability, followed by delivery method determination based on vascular access (Figure 10).

Subjects will be considered enrolled into the study after completion of all of the following steps:

- 1. Signed informed consent is obtained.
- 2. Based on the screening assessments, it is determined that the subject meets all of the inclusion and none of the exclusion criteria.
- 3. Subject is approved by the subject selection committee.
- 4. The trial cohort has been determined, and understood by the subject.
- 5. The subject is randomized (pivotal IDE only) or assigned to the appropriate registry or CAP.

In the FlexNav study and the CAP (under protocol version L), the subject will be considered enrolled once steps 1-4 above are complete and when the FlexNav™ Delivery System enters the subjects' body.

For the pivotal randomized IDE cohort, the subject will be randomized based on the cohort assignment as follows:

- The high risk cohort will be randomized against an FDA-approved and commercially-available transcatheter valve on a 1:1 basis.
- The extreme risk cohort will be randomized against an FDA-approved and commercially-available transcatheter valve on a 1:1 basis.

It is strongly recommended the implant procedure take place no later than 14 calendar days from subject enrollment/randomization

Once a subject is randomized in the pivotal IDE, crossover from one arm to the other is not allowed. However, following randomization or enrollment in the FlexNav Study, registry or the CAP, those subjects who are scheduled to receive a transcatheter valve via transfemoral access and found not to be suitable for this delivery modality (per the heart team medical decision) can receive a transcatheter valve using an alternate access modality and vice versa. However, this will be considered a protocol deviation unless multiple access routes were pre-approved by the Subject Selection Committee. The rationale for this decision must be documented.

In the pivotal IDE trial, when subjects are randomized to receive a CAV, the subject selection and procedure must follow the FDA-approved instructions for use (IFU).



TF=Transfemoral, CAV= FDA approved and commercially available transcatheter valve, AA=Alternative Access, V-in-V=Valve-in-Valve

**Figure 10. PORTICO Clinical Study Flow Chart** 

# 7 Study Conduct (Pivotal IDE and CAP)

# 7.1 Subject Informed Consent

Prior to enrolling in the clinical investigation, subjects shall be fully informed of the details of clinical investigation participation as required by applicable regulations and the center's IRB. Informed consent must be obtained from each subject prior to any clinical investigation participation (including the study-specific screening phase), using the Informed Consent Form (ICF). The ICF must be signed and dated by the subject and by the person obtaining the consent.

The subject shall be provided ample time to meet with the Site Principal Investigator or site personnel conducting the consent, and must be given the opportunity to ask questions of and receive satisfactory answers. The subject will then be allowed additional time, if requested, to take a copy of the informed consent form home with him or her to allow for additional time to thoroughly review this documentation.

All information pertinent to the clinical investigation shall be provided in writing and in native, non-technical language that is understandable to the subject.

The process of informed consent shall avoid any coercion of or undue influence of patients to participate, not waive or appear to waive patient's legal rights, use language that is non-technical and understandable to the patient, provide ample time for the patient to consider participation, and include dated signatures of the patient and of the clinical investigator or person obtaining the consent.

Prior to the subject signing the ICF, the Investigator or authorized delegate will fully explain to the subject the nature of the research, clinical investigation procedures, anticipated benefits, and potential risks of participation in the clinical investigation. The Investigator or delegate will allow adequate time for the subject to read and review the informed consent form and to ask questions.

The Investigator or authorized delegate must document in the subject's medical records that the subject was consented and the date on which the consent was obtained. The original signed informed consent form will be retained in the subject's clinical investigation records. A copy of the signed informed consent form and will be provided to the subject and a copy placed in the subject's medical record.

If new information becomes available during the clinical investigation that can significantly affect a subject's future health and medical care, or willingness to continue in the study, that information will be provided to the subject(s) in written form.

# 7.2 Subject Selection Committee

The Subject Selection Committee will be responsible for ensuring all subjects' clinical eligibility and technical suitability for implant according to the protocol. The composition and detailed process is further defined in the Subject Selection Committee Charter.

Subject Selection Committee review and approval is required prior to enrollment of any subject into any randomized cohort, FlexNav study, registry or the CAP.

#### 7.3 Index Procedure

The heart team's interventional cardiologist(s) and cardiac surgeon(s) must jointly participate in the intra-operative technical aspects of TAVR.

The index procedure should occur within 14 calendar days following subject randomization, registry or CAP assignment. The procedure must be performed according to the instructions for use (IFU) for the assigned device. Antiplatelet/Anticoagulation and other medications should be administered per the standard of care.

Cardiac enzymes must be obtained prior to the index procedure and within approximately 72 hours after the procedure.

Cardiac rhythm should be monitored and recorded at the following time points:

- 1. Upon crossing native valve with the guidewire
- 2. Upon positioning of the guidewire
- 3. Prior to valvuloplasty (if performed)
- 4. Immediately post valvuloplasty (if performed)
- 5. Before valve crosses the AV valve
- 6. After valve crosses the annulus
- 7. After valve is deployed in final position

The following data should be collected pre and post implant:

- Aortic systolic/diastolic pressure, Mean aortic pressure, Mean AV gradient, Peak AV gradient
- 2. Simultaneous Aortic and LV pressure measurements for valve area calculation
- 3. A supra-aortic angiogram for valve performance and coronary patency
- 4. Device deployment information
- 5. If performed, right atrial (RA) pressure, pulmonary artery (PA) systolic/diastolic pressure, Mean PA pressure, pulmonary wedge pressure (PCWP)

The activated clotting time (ACT) should be monitored and recorded on source documentation during the procedure and adjusted to attempt to keep the subject's ACT>250 seconds.

If an enrolled subject is not implanted with a TAVR valve, the following will apply:

- Randomized subjects will be followed per protocol through the one-year visit, as part of the primary analysis intent to treat (ITT) population, and then terminated from the study.
- Registry-assigned (Roll-in or Valve-in-Valve), FlexNav study and CAP subjects will be assessed for any adverse events through 30 days post procedure, and then terminated from the study.

#### **Post Procedure Activities**

- 1. Echocardiogram within 24-48 hours of procedure (or at discharge)
- 2. Troponin, or CK / CK-MB should be collected within approximately 12-24 hours after procedure, 24 hours thereafter, and at approximately 72 hours after the procedure (or at discharge, if patient is discharged prior to 72 hours post procedure)
- 3. BUN and Creatinine should be collected within 72 hours after index procedure

# 7.4 Discharge Visit (or up to 7 days post procedure, whichever occurs first)

The discharge visit will take place at the time of hospital discharge or up to 7 days after the procedure, whichever occurs first. If the subject is expected to be discharged over the weekend, the discharge tests may be completed on the last week day prior to discharge. The discharge assessment will include:

- 1. Physical exam
- 2. CCS Status of angina
- 3. Modified Rankin Scale (mRS)
- 4. NIH Stroke Scale (NIHSS)
- 5. Barthel Index
- 6. Echocardiogram (if not performed during the post procedure testing within 24-48 hours after procedure)
- 7. 12 lead ECG (for subjects receiving a new permanent pacemaker, ECG should be completed showing the underlying rhythm as well as the current pacing programming)
- 8. Cardiovascular medications documentation
- 9. Adverse events assessment
- 10. Lab Measurements (per Table 9, Table of Assessments)

# 7.5 Follow-up Visits

Every effort should be made by the study site to have the subject return to the investigative center for all study visits. If, despite all efforts, the subject is unable to return to the study site in-person during a follow-up window, subjects may undergo a remote follow-up assessment to collect applicable data. Remote assessments should include all data that can be reasonably and legally collected remotely on the study subject. Visits occurring at non-study sites will be limited to standard of care data collection. Authorization for the release of medical records from non-study facility is the responsibility of the study site. Protocol deviations will be required for all missed testing.

# 7.6 30 Day Visit (±7 days)

The 30 Day visit will take place 30 days (±7 days) post index procedure, and will include the following:

- Physical exam
- 2. CCS status of angina
- 3. Modified Rankin Scale (mRS)
- 4. NIH Stroke Scale (NIHSS)
- 5. Barthel Index
- 6. Echocardiography
- 7. 12 lead ECG (for subjects receiving a new permanent pacemaker, ECG should be completed showing the underlying rhythm as well as the current pacing programming)
- 8. Lab Measurements (per Table 9, Table of Assessments)
- 9. NYHA Functional Classification
- 10. Frailty Index assessment
- 11. Quality of Life Measures (For CAP subjects enrolled under Ver. K or later, only the KCCQ and EQ-5D are required.)
- 12. MMSE-2:SV
- 13. Six Minute Walk Test (6MWT) (Not required for CAP subjects enrolled under Ver. K or later)
- 14. Cardiovascular medications
- 15. Adverse events assessment
- 16. Multi-Slice CT (MSCT) Scan (or TEE if MSCT is medically or technically contraindicated), as described in Appendix S: TAVR Leaflet Motion Sub-study until sub-study enrollment is complete. (Not required for subjects enrolled under Ver. K or later)

# 7.7 6 Month (±30 days) (This visit is not required for CAP subjects enrolled under Ver. K or later)

The following data must be collected at 6 Months post index procedure:

- 1. Physical exam
- 2. CCS status of angina
- 3. Modified Rankin Scale (mRS)
- 4. NIH Stroke Scale (NIHSS)
- 5. Barthel Index
- 6. Echocardiography
- 12 lead ECG (for subjects receiving a new permanent pacemaker, ECG should be completed showing the underlying rhythm as well as the current pacing programming)
- 8. Lab Measurements (per Table 9, Table of Assessments)
- 9. NYHA Functional Classification
- 10. Frailty Index assessment
- 11. Quality of Life Measures (QoL)
- 12. MMSE-2:SV

- 13. Six Minute Walk Test (6MWT)
- 14. Cardiovascular medications
- 15. Adverse events assessment

  Multi-Slice CT (MSCT) Scan (or TEE if MSCT is medically or technically
  contraindicated), as described in Appendix S: TAVR Leaflet Motion Sub-study
  until sub-study enrollment is complete.

# 7.8 One-Year Visit (-30 days, + 45 days)

The following data must be collected at one-year (-30 days, + 45 days) post index procedure:

- 1. Physical exam
- 2. CCS status of angina
- 3. Modified Rankin Scale (mRS)
- 4. NIH Stroke Scale (NIHSS)
- 5. Barthel Index
- 6. Echocardiography
- 7. 12 lead ECG (for subjects receiving a new permanent pacemaker, ECG should be completed showing the underlying rhythm as well as the current pacing programming)
- 8. Lab Measurements (per Table 9, Table of Assessments)
- 9. NYHA Functional Classification
- 10. Frailty Index assessment
- 11. Quality of Life Measures (QoL) (For CAP subjects enrolled under Ver. K or later, only the KCCQ and EQ-5D are required.)
- 12. MMSE-2:SV
- 13. Six Minute Walk Test (6MWT) (Not required for CAP subjects enrolled under Ver. K or later)
- 14. Cardiovascular medications documentation
- 15. Adverse events assessment

# 7.9 Annual Visits (2 year, 3 year, 4 year and 5 year (±60 days))

The following data should be collected at years 2, 3, 4 and 5 post index procedure:

- 1. Physical exam
- 2. CCS status of angina
- 3. NYHA Functional Classification
- 4. Cardiovascular medications
- 5. Adverse event assessment
- 6. NIH Stroke Scale (NIHSS)
- 7. Modified Rankin Stroke Scale
- 8. Barthel Index

- 12 lead ECG (for subjects receiving a new permanent pacemaker, ECG should be completed showing the underlying rhythm as well as the current pacing programming)
- 10. Echocardiography
- 11. Quality of Life Measures (QoL) (For CAP subjects enrolled under Ver. K or later, only the KCCQ and EQ-5D are required.)

#### 7.10 Unscheduled Visits

# 7.10.1 Unscheduled Visits for Evaluation of Suspected Neurological Event

If the subject experiences a neurological event (TIA, stroke, or encephalopathy), the event should be documented on an adverse event form and further evaluation should be performed at an unscheduled visit 90 days\* (±14 days) from the date of the neurological event. The unscheduled visit will include the following assessments:

- 1. Neurological Assessment conducted by a neurologist or a neurology fellow
- 2. NIH Stroke Scale
- 3. Modified Rankin Scale (mRS)

# 7.11 Evaluation of Ischemic Stroke and Myocardial Infarction

All ischemic strokes and myocardial infarctions should be investigated per standard of care to include an assessment for leaflet motion (TEE is recommended) and evaluation of sources for an embolus (e.g., left atrial appendage).

#### 7.12 Subject Withdrawal

All living and enrolled subjects are required to complete clinical follow-up. A study subject that has been withdrawn from the study will not be replaced. All data collected up to the point of their study discontinuation will be reported and included in the data analysis as applicable.

If a subject cannot be reached for a follow-up visit, the investigator will complete a Protocol Deviation Case Report Form. The efforts undertaken to contact the subject, referring physicians, including internists as well as cardiologists, family members, or other alternate contacts should be noted in the subject's records. These efforts should include at least three (3) attempts of telephone contact on separate dates, and a registered letter before considering the subject lost-to-follow-up.

#### 7.13 Table of Assessments

Subject data and data collection timeline are summarized in Table 9.

<sup>\*</sup> FDA's Current Thinking Regarding Neurological Assessments for Transcatheter Valve Trials (Revised: August 25, 2011)

Table 9. Table of Assessments (IDE Pivotal Trial and CAP)





# **7.14 Study Activity Definitions**

Table 10 summarizes the study activity definitions.

| Charles A skinds | Definition. |
|---|---|
| Study Activity | Definition |
| Adverse Event<br>Assessment | All adverse events will be documented according to Adverse Events section 9. |
| Lab Measurements | The following lab tests will be collected at each required interval per Table 9, Table of Assessments: |
| Barthel Index | A scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility where a higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from the hospital. |
| Cardiac Rhythm | Assessment of heart rate, QRS and dominant rhythm pre-procedure, during |
| Monitoring | and after the procedure. |
| CCS Angina | Canadian Cardiovascular Society grading of angina pectoris (Appendix I) |
| Coronary and Aortic<br>Angiogram (with runoff<br>if clinically indicated) | Coronary and aortic imaging conducted per institutional guidelines. |
| CT Scan/MSCT Scan | Computed Tomography (CT) with minimum of 64-detectors is recommended for image acquisition. The complete cardiac cycle will be captured, encompassing both the diastolic and systolic phases of the heart (Multi-Slice). Scan records that leave the institution will be modified to remove subject identifiers. CT Scan images will be provided to a CT core lab for evaluation. |
| Echocardiography | Each site is responsible for performing the echocardiogram according to the Echocardiographic protocol. Echocardiogram will be provided to an Echocardiographic core lab for evaluation. |
| 12 lead<br>Electrocardiogram (ECG) | Assessment of heart rate, QRS and dominant rhythm using 12 lead ECG. For subjects receiving a permanent pacemaker during the study, an ECG will be completed showing the underlying rhythm as well as the current pacing programming. Electrocardiograms will be provided to an Electrocardiographic core lab for evaluation. |
| FEV1 | The volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. |
| Frailty Index | Used to assess if frailty is a high risk factor for subjects prior to enrollment. |
| Informed Consent | An IRB- and Sponsor-approved Informed Consent must be obtained before subject enrollment |
| Medical History | General medical history of the subject: |

| Cardiovascular<br>Medications | <ul> <li>Previous cardiovascular operations</li> <li>Coexisting cardiovascular diseases</li> <li>Clinically significant peripheral vascular disease (PVD)</li> <li>Previous peripheral vascular operations</li> <li>Other coexisting medical conditions (e.g., diabetes, hypertension, kidney and lung disease, endocarditis)</li> <li>Only the following Cardiovascular medications will be collected at each visit: <ul> <li>Beta Blockers</li> </ul> </li> <li>Calcium Channel Blockers</li> <li>Anticoagulants</li> <li>Antiplatelet agents including Aspirin</li> <li>Diuretics</li> <li>Ace-Inhibitors</li> <li>Angiotensin Receptor Blocker (ARBs)</li> <li>Hydralazine</li> </ul> |
|---|---|
| | Antiarrhythmics |
| MMSE-2:SV | Mini Mental State Exam -2:SV is a screening tool for cognitive impairment |
| Modified Rankin Stroke<br>Scale* | The modified Rankin Scale (mRS) is functional measurement to assess the degree of disability or dependence in the daily activities of people who have suffered a stroke. *This assessment must be completed by a rater who has a current certificate that demonstrates completion of an accredited training program for this stroke scale, or by a neurologist or neurology fellow. |
| Multidisciplinary Heart<br>Team | All suitable subjects must undergo the established institutional specific multidisciplinary/Heart team (as defined in the CMS Decision Memo for TAVR (CAG-00430N) assessment to confirm both appropriateness for transcatheter aortic valve placement and high-risk designation. Both co- investigators must be involved in the subject selection and screening process. All subjects evaluated for severe aortic stenosis in medical and surgical departments that are high or extreme risk candidates for AVR should be screened for study eligibility. |
| Neurological Assessment | A neurological assessment will be conducted on subjects 90 days (±14 days) after any neurological event (stroke, TIA, encephalopathy). The neurological assessment should be conducted by a <b>neurologist or a neurology fellow</b> and should include physical functioning as well as a basic neurocognitive evaluation to cover the major domains. |
| NIH Stroke Scale** | The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Certified personnel rate the subject's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single subject assessment requires less than 10 minutes to complete. |
| | ** National Institute of Health (NIH) Stroke Scale - All personnel conducting any study required NIHSS evaluations are required to have received training and certification per nationally accepted guidelines such as American Stroke Association, or American Academy of Neurology, or National Institute of |

| | Neurological Disorders and Stroke, or must be a neurologist or neurology |
|---|---|
| | fellow. |
| NYHA Classification | The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying the extent of heart failure. It places subjects in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regards to normal breathing and varying degrees in shortness of breath and or angina pain |
| Physical Assessment | At the baseline visit the following measurement must be assessed: |
| Procedure Information | <ul> <li>Procedure information must be collected including:</li> <li>Pre-procedure Information</li> <li>Procedure Information</li> <li>Post-procedure Information</li> </ul> |
| Quality of Life Measures | EQ-5D 3L is a standardized instrument for use as a measure of health outcomes. The process to complete this questionnaire is indicated. SF-36 is a survey of subject health to determine cost-effectiveness of a health treatment KCCQ is a 23 item questionnaire that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life |
| Surgical Risk Assessment | Surgical Risk Assessment tools consist of EuroSCORE II and STS Risk Score. |
| Six Minute Walk Test | The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. |
| Subject Selection<br>Committee | The Subject Selection Committee will be responsible for ensuring all subjects' clinical eligibility and technical suitability for implant according to the protocol. The composition and detailed process is further defined in the Subject Selection Committee Charter. |

# 7.15 Determination of the Aortic Annulus Size

The PORTICO clinical study requires that all annulus sizing be determined using a CT scan for all participants in the study. However, if CT is contraindicated and/or not possible to be obtained for certain subjects, a 3D echocardiogram and non-contrast CT of chest and abdomen/pelvis may be accepted if approved by the Subject Selection Committee.

#### 7.16 Core Laboratories

Independent core laboratories will be utilized for evaluating CT images, ECG rhythms and echocardiograms for the pivotal IDE cohort. The same core laboratories and processes will be used for the CT images and echocardiograms for the CAP cohort.

Each site is responsible for performing the CT scan and echocardiogram according to the core laboratory imaging protocol. Also, ECG data collection and reporting must be completed according to the ECG core laboratory protocol.

CT scan, echocardiography, and ECG data will be forwarded to the respective core laboratories for interpretation. It is the responsibility of each site to perform the local interpretation of the echocardiogram for clinical assessment.

The core laboratories will not be responsible for notifying the site of any abnormal findings that are identified in the study. The responsibility of the core laboratories is to complete the data collection forms and submit these to the Sponsor.

The core laboratories will provide the study required interpretation and documentation of each data submission. Data obtained from the core laboratory readings will be used for study purposes only and not for clinical treatment of the subject. The Sponsor will use only the measurements provided by the core laboratories in data analyses. If the core laboratory determines that the data are unreadable, the site will be responsible for having the subject return for another assessment.

# 7.17 Medications

If a subject is taking any of the following classes of cardiovascular medications, they will be reviewed at each applicable visit and documented on the visit CRF:

- Beta Blockers
- 2. Calcium Channel Blockers
- 3. Anticoagulants
- 4. Antiplatelet agents including Aspirin
- 5. Diuretics
- 6. Ace-Inhibitors
- 7. Angiotensin Receptor Blocker (ARBs)
- 8. Hydralazine
- 9. Antiarrhythmics

# 8 Data Collection and Management (Pivotal IDE and CAP)

A study-specific Data Management Plan will be created to document measures ensuring data quality and completeness. All required study data will be recorded on study-specific electronic Case Report Forms (eCRFs), as provided by SJM.

Subject data will be collected using a web-based remote electronic data capture (EDC/RDC) system supported by SJM. The Investigator or his/her designee is responsible for timely recording of all data onto the study eCRFs. The data used to complete these forms has to be verified by authorized site personnel.

If additional documentation (e.g., procedural notes, discharge summaries) is required for any reason (such as an adverse event) it should be appropriately redacted (e.g., blacked out) to remove the subject's name and any additional identifying information, and the subject's unique study ID code inserted, prior to being submitted to SJM.

# 8.1 Source Data and Subject Files

The Investigator has to keep a written or electronic subject file for every subject participating in the clinical study. In this subject file, the available demographic and medical information of a subject has to be documented, in particular the following:

- 1. Name
- 2. Birth date
- 3. Sex
- 4. Height
- 5. Weight
- 6. Ethnicity (if available)
- 7. Medical history
- 8. Concomitant diseases and concomitant medications (including changes during the course of the study)
- 9. Statement of entry into the study
- 10. Study identification
- 11. Date of informed consent
- 12. All study visit dates
- 13. Predefined performed examinations and clinical findings
- 14. Observed AEs and source documents related to the AE
- 15. Reason for withdrawal from the study, if applicable.

It should be possible to verify the inclusion and exclusion criteria for the study from the available data in this file.

It must be possible for the investigator to identify each subject by using this subject file.

Additionally, any other documents with source data that were generated by technical equipment have to be filed. This may include 12 lead ECG recordings, X-ray films, CT scans and laboratory value listings, as applicable. All these documents have to bear at least the subject identification. The medical evaluation of such records should be

documented as necessary. All data recorded on the eCRF must be found in the subject's source data.



# 9 Adverse Events (Pivotal IDE and CAP)

# 9.1 Unanticipated Adverse Device Effect

Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application, including a supplementary plan or application, or any other unanticipated serious problem associated with the device that relates to the rights, safety, or welfare of subjects (21 CFR 812.3 (s)).

# 9.2 Anticipated Adverse Events

Adverse Events will be classified as either a Serious Adverse Event or an Adverse Event.

**Serious Adverse Event**- is defined as those adverse events resulting in the following: death, life-threatening adverse event, unplanned inpatient hospitalization or prolongation of existing hospital stay, persistent or significant disability/incapacity, congenital anomaly/birth defect or medically significant event.

**Adverse Event** - is defined as an event which does not meet the definition of a serious adverse event but is still an undesirable clinical occurrence and is a negative change from baseline, whether or not device related

# 9.3 Potential Anticipated Adverse Events

The potential anticipated adverse events include but are not limited to, the following:

- 1. Access site complications (e.g., pain, bleeding, infection, hematoma, pseudoaneurysm, etc.)
- 2. Acute coronary obstruction
- 3. Acute myocardial infarction
- 4. Access site injury
- 5. Allergic reaction to antiplatelet agents, contrast medium, anesthesia, or valve components
- 6. Anaphylactic shock/toxic reaction
- 7. Annulus rupture
- 8. Aortic rupture
- 9. Ascending aorta trauma
- 10. Atrio-ventricular node block
- 11. AV fistula
- 12. Bleeding
- 13. Cardiac arrhythmias
- 14. Cardiovascular or vascular injury, such as perforation or damage (dissection) of vessels, ventricle, myocardium or valvular structures that may require intervention
- 15. Conduction system injury
- 16. Death

- 17. Endocarditis
- 18. Embolism: air, calcification or thrombus
- 19. Exercise intolerance (weakness)
- 20. Fever
- 21. Heart failure
- 22. Hematoma
- 23. Hemodynamic compromise
- 24. Hemolysis
- 25. Hemolytic anemia
- 26. Hemorrhage
- 27. Hypotension or hypertension
- 28. Immunological reaction
- 29. Infection
- 30. Leakage, regurgitation
- 31. Left ventricular failure/rupture
- 32. Left ventricular impairment (due to apical scar)
- 33. Myocardial ischemia
- 34. Mitral valve insufficiency
- 35. Multi-organ failure
- 36. Neurological changes including stroke/transient ischemic attack;
- 37. Non-structural dysfunction (i.e., entrapment by pannus, paravalvular leak, inappropriate sizing or positioning)
- 38. Pannus
- 39. Paravalvular leak
- 40. Pericardial effusion
- 41. Perforation of the myocardium or a blood vessel
- 42. Potential coronary obstruction
- 43. Renal failure
- 44. Renal insufficiency
- 45. Respiratory failure (shortness of breath)
- 46. Sepsis
- 47. Septal rupture
- 48. Stenosis (high gradient)
- 49. Stroke
- 50. Structural valve deterioration (i.e., calcification, leaflet tear)
- 51. Systemic peripheral ischemia
- 52. Tamponade
- 53. Valve explant
- 54. Valve embolization
- 55. Valve migration or malposition
- 56. Valve stenosis
- 57. Valve thrombosis
- 58. Ventricular failure (acute)
- 59. Ventricular rupture

# 60. Vessel dissection or spasm

It is possible these complications could lead to:

- 1. Transfusion
- 2. Conversion to open surgical procedure
- 3. Reoperation
- 4. Emergent balloon valvuloplasty
- 5. Emergent percutaneous coronary intervention (PCI)
- 6. Emergent surgery (i.e., coronary artery bypass, heart valve replacement)
- 7. Explantation
- 8. Permanent disability
- 9. Death
- 10. Permanent pacemaker

There are no known interactions of the Portico Transcatheter Heart Valve with concomitant medical treatment.

Subjects experiencing an adverse event shall be treated per the standard of care at the investigation site.

# 9.4 Adverse Event Reporting

# 9.4.1 Reporting All Adverse Events

Investigators are responsible for promptly reporting ALL adverse events to SJM by completing the Adverse Event eCRF. Serious Adverse Events must be reported to the Sponsor no later than three (3) calendar days from the day the site personnel became aware of the event or as per the investigative site's local requirements, if the requirement is more stringent than those outlined above. All unresolved adverse events should be followed by the investigator until resolution.

For subjects enrolled under version L or later of the protocol, the reporting of adverse events will commence at the time of the Portico implant attempt.

# 9.4.2 Paravalvular Leak

Paravalvular leak should be reported as an adverse event in the following cases:

- When paravalvular leak remains moderate or severe after balloon dilatation, or
- When valve-in-valve, surgical conversion or other intervention is required for any grade of paravalvular leak after implant.

# 9.4.3 Reporting Unanticipated Adverse Device Effects

An investigator shall submit to the Sponsor and the reviewing IRB a report of any unanticipated adverse device effect occurring during an investigation no later than three (3) calendar days from the day the site personnel first learns of the effect.

#### 9.5 Classification of Causal Relationships

For each adverse event, the causal relationship between the adverse event and the Portico Transcatheter Heart Valve and Delivery System, and the causal relationship between the event and the index procedure, will be assessed by the Investigator and reported as such on the Adverse Event case report form. Final causal relationships for events related to primary and secondary endpoint criteria according to the Valve Academic Research Consortium (VARC 2) definitions will be determined per CEC adjudication.

#### 9.6 Subject Death

Subject death is a potential outcome of a Serious Adverse Event that will be reported within three (3) calendar days from the time of the site personnel knowledge of the event, if the event occurs from the time of signed informed consent until the subject exits the study.

Subject death will be subdivided specifically denoting cardiovascular and non-cardiovascular mortality:

- 1. Cardiovascular mortality includes any one of the following criteria:
  - a. Any death due to proximate cardiac cause (such as MI, tamponade, worsening heart failure)
  - b. Sudden or unwitnessed death
  - c. Death of unknown cause
  - d. All procedure-related deaths including those related to a complication of the procedure or treatment for a complication of the procedure
  - e. Death caused by non-coronary vascular conditions such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular disease.
- 2. Non-cardiovascular mortality includes any death in which the primary cause of death is clearly related to another condition (e.g. trauma, cancer, suicide)

An Adverse Event CRF, Death CRF and relevant source documentation including the death certificate should be submitted to SJM.

#### 10 Independent Boards (Pivotal IDE and CAP)

#### 10.1 Clinical Events Committee

An independent Clinical Events Committee (CEC), consisting of, at a minimum, an interventional cardiologist, cardiologist, cardiothoracic surgeon, and a neurologist will adjudicate events related to primary and secondary endpoint criteria according to the Valve Academic Research Consortium (VARC 2) definitions. The CEC will have final adjudication responsibilities for subject outcomes related to primary and secondary endpoint criteria. Members of the CEC cannot be investigators on the PORTICO Clinical

Study. A charter that is agreed upon by both the Sponsor and the independent CEC governs the event adjudication process.

# 10.2 Data Safety Monitoring Board (DSMB) (Pivotal IDE)

An independent Data Safety Monitoring Board (DSMB) will be utilized to regularly review study progress with regard to safety of the pivotal IDE trial. Members of the DSMB cannot be investigators on the PORTICO Clinical Study. Board membership may consist of, but not limited to, a cardiologist, cardiac surgeon, neurologists, and a biostatistician.

The primary responsibilities of the DSMB include:

- Review and validate the subject sample (i.e., review inclusion/exclusion deviations and other protocol deviations)
- Provide oversight for issues affecting general subject welfare
- Recommend premature study termination or modification of the trial for any perceived safety concerns

At any time during the course of the study, the DSMB may offer opinions or make formal recommendations concerning aspects of the study that impact subject safety (e.g., safety-related protocol changes or input regarding adverse event rates associated with the investigational study). Additionally, the DSMB may act as an advisory panel for questions regarding informed consent, subject enrollment, protocol implementation, study endpoints, data discrepancies, and other issues that may present during the course of the study. A charter that is agreed upon by both the sponsor and the DSMB members governs the role and responsibility of this committee.

The recommendations of the DSMB are not binding, and all final decisions related to modifications to the clinical investigational protocol rest with the Sponsor.

# 11 Statistical Methods and Analysis (Pivotal IDE)

This section describes the statistical methods and analysis of the pivotal IDE randomized cohort unless otherwise specified. The analysis will be performed on combined high-risk cohort and extreme-risk cohort.

# 11.1 Analysis Populations

The primary analysis will be based on the intention-to-treat (ITT) population. The ITT population is defined

Additional populations will be used to confirm the results of the ITT population.



# 11.2 Randomization and Stratification



# 11.3 Primary Endpoints

# 11.3.1 Primary Effectiveness Endpoint

The primary effectiveness endpoint is the composite endpoint of all-cause mortality or disabling stroke at one year. This endpoint will be evaluated by a non-inferiority test comparing the Portico test group to the control (CAV) group, and the primary analysis will be conducted on the ITT population.





# 11.3.2 Primary Safety Endpoint

The primary safety endpoint is the non-hierarchical composite endpoint of all-cause mortality, disabling stroke, life-threatening bleeding requiring blood transfusion, acute kidney injury requiring dialysis, or major vascular complications at 30 days. This endpoint will be evaluated by a non-inferiority test comparing Portico test group to the control group, and the primary analysis will be conducted on the ITT population.





# 11.4.1 Sample Size for the Primary Effectiveness Endpoint





# 11.4.2 Sample Size for the Primary Safety Endpoint



# 11.4.3 Total Sample Size

The total sample size required for evaluating the primary effectiveness and safety endpoints is 750 and 750 subjects respectively. Thus the total sample size is 750 for the study.



# 11.5 Secondary Endpoints

All secondary endpoints are defined in section 1.3. Among these, 4 have hypotheses to be tested. The secondary study hypotheses are:

- Severe aortic regurgitation (AR) at one year
- Kansas City Cardiomyopathy Questionnaire (KCCQ) at one year
- Moderate or severe aortic regurgitation at one year

• 6-minute walk at one year Non-inferiority tests will be performed for each endpoint.










# 11.7.4 Analysis of Descriptive Endpoints

The descriptive endpoints listed in section 1.3 will be summarized using descriptive statistics including mean, standard deviation, median and range for continuous data and count and percentage for categorical data.


### 11.10 Statistical Methods and Analysis (FlexNav Study, Registries and CAP)



### 12 Study Termination/Withdrawal (Pivotal IDE and CAP)

Active subject participation in the pivotal IDE is expected to last for five (5) years after index procedure unless the subject was randomized or assigned to a registry or FlexNav study but not implanted with a TAVR valve. Enrolled CAP subjects successfully implanted with a Portico valve will be followed for a minimum of one year and up to 5 years or upon study completion (whichever is reached first).

If an enrolled subject was not implanted with a TAVR valve, the following will apply:

- Randomized subjects will be followed per protocol through to the one-year visit, as part of the primary analysis intent to treat (ITT) population, and then terminated from the study.
- Registry-assigned (Roll-in or VIV Registry), FlexNav study or CAP subjects will be assessed for any adverse events through 30 days post procedure, and then terminated from the study.

The study will be closed at the investigational site following the distribution of the final clinical study report for all study locations. A copy of the final report will be provided to the IRB and Competent Authorities, if applicable, and acknowledgement requested.

Early termination of the study by either SJM or the Investigator, if applicable, will be communicated to the IRB.

Upon completion of subject participation in this study, the subject will be followed-up in accordance with institutional standards.

Possible reasons for early termination of the study and/or investigation site's participation in the study may include, but are not limited to:

- Request from the Clinical Investigation Site Principal Investigator
- Delivery system or device fails to perform as intended
- Occurrence of UADE which cannot be prevented in future cases
- SJM management decision to discontinue the study

- Request from Regulatory bodies
- Site's noncompliance with the requirements of the CIP and/or applicable laws and regulations
- Falsification of data or any other breach of ethics or scientific principles

Subjects must be informed about their right to withdraw from the study at any time and for any reason without sanction, penalty, or loss of benefits to which the subject is otherwise entitled and withdrawal from the study will not jeopardize their future medical care or their relationship with the Principal Investigator. Subjects will be asked what the reason for termination is but have the right not to answer.

The Principal Investigator may withdraw a subject from the study at any time if s/he believes it is in the subject's best interest.

The subject's future care will not be changed by a decision, voluntary or otherwise, to withdraw from the study. All reasonable efforts should be made to retain the subject in the clinical study until completion of the clinical study.

Reasons for subject's termination or withdrawal include, but are not limited to, the following:

- Subject death (in case of subject death, cause must be documented)
- Subject and/or family request, if applicable
- Subject non-compliance
- Subject lost to follow-up, defined as the following: a subject will be considered "lost to follow-up" after a minimum of 3 documented phone calls of a physician or designee at the study site to the subject or emergency contact and a letter sent to the last known address
- Subject's participation terminated by the Principal Investigator
- Study discontinued due to management decision by sponsor or request from Regulatory bodies
- Investigational site ends participation in the study

The study will be terminated according to locally applicable regulations. If applicable, the study may be temporarily suspended or terminated, either at the local, national, or international level, at the request of the IRB and/or the FDA. Justification and request for resuming the clinical investigation after suspension will be communicated to the IRB and the FDA.

### 13 Study Management (Pivotal IDE and CAP)

SJM, as the study sponsor, is responsible for:

- the design, overall conduct, analysis, and reporting of the results from this study as described in this CIP
- conducting CIP and technical training of the Principal Investigator and Co-Investigator(s)
- conducting CIP training of clinical staff, including but not limited to, research coordinator(s), echocardiographers, procedural staff
- monitoring the study
- performing those actions necessary to protect the rights of subjects and the scientific credibility of this study is conducted
- selecting qualified study Investigators, study monitors and research staff
- safety reporting to Competent Authorities
- providing support from a Field Clinical Specialist at each Portico valve implant
- providing a proctor as support for each Portico valve implant until the proctor/SJM determines the site can function independently

SJM reserves the right to obtain data clarification and/or additional medical documentation on subjects enrolled in this study until the study is terminated or closed by study final report.

The Sponsor of this study and manufacturer of the investigational device is:



SJM will retain, at a minimum, the following reports, records, publications:

- Signed Clinical Investigation Plan and all amendments
- Blank, revision controlled eCRFs
- Informed Consent Form template, and all IRB-approved versions
- Signed Study Agreements and all amendments completed
- Investigator Financial Disclosure information and all updates thereto
- IRB approval letters
- Regulatory approval letters
- All significant correspondence relating to the conduct of this study between SJM the study site, and IRB
- Signed CVs and professional licenses (if applicable) for all study personnel
- Training records relevant to conduct of the Clinical Investigation
- CIP/device related training records for all applicable study personnel

- Site personnel signatures and documentation of the Investigator's delegation of study related responsibilities
- Investigational device inventory information including the date, quantity, and unique identifier of all investigational devices shipped and received
- Appropriate tracking of each investigational device to include implant, explant, return, and analysis
- Publication Agreement
- IRB Registration Number
- List of IRB voting members (optional)
- Insurance Certificate
- Relevant Source Documentation (de-identified).

## **13.1** Study Investigators

Study Investigators are those who have been qualified and sufficiently trained by SJM on the study CIP requirements. Implanting Study Investigators have to complete required training as per the Training Plan prior to implanting the Portico Transcatheter Heart Valve.

### **13.2** National Principal Investigators



### 13.3 Investigator Responsibilities







## 13.5 Records



# 13.6 Record Retention





### 13.7 Confidentiality

All subject information collected during the course of this study will be kept strictly confidential according to applicable country-specific laws and regulations. All data and information concerning subjects and their participation in this study are considered confidential by Sponsor, and its affiliates (located in the U.S.A. and European Economic Area (EEA), and other countries), and other people who work for Sponsor to provide services related to the device and this study (collectively referred to as "SJM"). All public reporting of the results of the study will eliminate identifiable references to the subjects. Information on paper will be kept in secured locations. Electronic information will be kept on password-protected computers.



Study subjects have a right to gain access and to correct inaccuracies in information about them as permitted by applicable law. In order to help keep subject medical records and personal information confidential only certain authorized investigators and sponsor personnel, or approved contracted agents of the sponsor, will have access to confidential records. These include researchers in the hospital who are part of this study, the sponsor and its affiliates and representatives that perform study-related services who may be located in the USA, European Economic Area (EEA) and other countries. The IRB and other regulatory authorities also have the right to inspect and copy records pertinent to this study. It is necessary for them to review study data, portions of study subject records and information so that they can follow the study progress, which may include without limitation:

- 1. monitor the accuracy and completeness of the study
- 2. perform scientific analysis and develop the medical product
- 3. and/or obtain approval to market the medical products in the USA, Canada, EEA, and other countries.

Any information about subjects that leaves the institution conducting the study will be modified to remove certain information that could identify the subject (e.g., subject's name, address, and hospital number) and only be identifiable by a study ID code. Study data provided to sponsor that is published in medical journals and/or presented at scientific conferences will not allow the identification of study subjects.

The results of the study will be made available to the sponsor and its affiliates (located in the U.S.A., EEA, and other countries) along with other people who work for the sponsor to provide services related to the device and this study and study center.

A summary of the information on all subjects may be provided to governmental agencies (including regulatory agencies), regulatory authorities in the U.S.A., Canada, EEA and other countries who may also need to review study data and portions of medical records. Results from this study may also be published in scientific journals or presented at conferences as an oral or poster presentation; however, the identity of a study subject will not be disclosed.

### 13.8 Amendment Procedure

If an amendment becomes necessary during the study, the site along with SJM will submit the CIP amendment to the IRB. SJM will submit the amendment to the FDA, as required. Prior approval from the FDA and IRB will need to be obtained, when applicable, prior to the implementation of the change except in an emergency situation to protect the health and welfare of the subject(s) as deemed necessary by the Principal Investigator.

A justification statement shall be included with each amended section of the CIP documentation, and the version number and dates of amendments will be documented.

### 13.9 Ethical Basis

The PORTICO clinical study will be performed in compliance with all applicable Federal regulations concerning the protection of human subjects found in the Code of Federal Regulations (CFR) and 21 CFR Parts 50 and 56.

This clinical investigation will be performed in accordance with the World Medical Association Declaration of Helsinki and 21 CFR parts 54 and 812.

IRB approval letter should clearly identify:

- the date of the meeting
- duration of approval or expiration date of approval
- the approved version of the Clinical Investigation Plan
- the approved version of the informed consent form and any other advertising or subject recruitment materials
- the approved version of the Instructions for Use (IFU)

Approval from the IRB is necessary prior to the start of the investigation. The original approval is to be filed in the Investigator Study Binder and a copy of the approval is provided to SJM prior to the first investigational assessment.

Any amendments to the CIP should be submitted to the FDA. Approval of amendments shall be obtained in written form from the FDA and IRB prior to implementation.

The IRB will be informed about SAEs, UADEs, and protocol deviations in accordance with local and national requirements.

### 13.10 Insurance

Subjects will be allowed to participate in the study regardless of their personal health insurance status.

### 13.11 Subpopulations

The PORTICO clinical study will include study patients with severe, symptomatic aortic stenosis that can be considered as one of three subpopulations:

- High operative risk for surgical aortic valve replacement
- Extreme operative risk for surgical aortic valve replacement
- Patients at either high or extreme operative risk who will have a TAVR valve implanted in an existing failed bioprosthetic surgical aortic valve.

### **13.12 Underrepresented Group Considerations**

Since findings based on data collected from trials are commonly used to support the application of therapies across the general population, it is important that the enrolled patient population be as representative as possible of the eligible population in terms of the racial, ethnic and gender mix.

The PORTICO clinical study inclusion and exclusion criteria do not unduly exclude any particular underrepresented group. In order to facilitate access to the study by underrepresented groups, the PORTICO clinical study will be conducted at sites throughout the United States and Australia and will consist of urban as well as rural facilities. Steps (e.g., translation of ICF to native language, financial hardship program, etc.) will be taken to ensure inclusion of underrepresented groups.

### 13.13 Study Monitoring

Investigational sites will be monitored to ensure the study is being conducted in accordance with this Clinical Investigation Plan, Investigator Agreement, applicable laws and regulations and SJM policies and procedures. Qualified clinical representatives will be selected to monitor this study. If required, a study-specific Monitoring Plan will be created. The Monitoring Plan will be in accordance with SJM procedures and will be updated as appropriate.



### 13.14 Regulatory Inspections

The Investigator and/or designee should contact SJM immediately upon notification of an impending FDA inspection.

An Investigator who has authority to grant access shall permit authorized FDA employees, at reasonable times and in reasonable manner, to enter and inspect any establishment where devices are held (including any establishment where devices are used or where records or results are kept).

An Investigator, or designee, shall permit authorized FDA employees, at reasonable times and in a reasonable manner, to inspect and copy all records relating to an investigation.

An Investigator shall permit authorized FDA employees to inspect and copy records that identify subjects, upon notice that FDA has reason to suspect that adequate informed consent was not obtained, or that reports required to be submitted by the investigator,

to the sponsor or IRB have not been submitted or are incomplete, inaccurate, false, or misleading.



### 13.16 Protocol Deviation

The Principal Investigator and delegates are required to adhere to the Clinical Investigation Plan, signed Study Agreement, applicable national or local laws and regulations, and any conditions required by the reviewing IRB or applicable regulatory authorities.

A protocol deviation is used to describe situations in which the CIP was not followed. All deviations must be reported to SJM on the Protocol Deviation Case Report Form. Deviations must be reported to the IRB per their requirements. Any corrective and preventive actions required by the IRB must be completed by the site.

The Investigator must notify SJM and the IRB (as required by the IRB's requirements) of any deviation from the Investigation Plan to protect the life or physical well-being of a subject in an emergency as soon as possible, but no later than 5 working days after the deviation has occurred.

SJM retains the right to terminate the participation of a study Investigator for any of, but not limited to, the following reasons:

- Concern for subject safety and welfare
- Failure to secure informed consent prior to any study activity
- Failure to report unanticipated adverse device effects without unjustified delay
- Repeated non-compliance with this Investigation Plan or the Study Agreement
- Inability to successfully implement this Investigation Plan
- Violation of the Declaration of Helsinki
- Violation of applicable national or local laws and regulations
- Falsification of data, or any other breach of ethics or scientific principles
- Loss of or unaccounted use of investigational device inventory
- Management decision by SJM

### 13.17 Device Accountability

The study site must maintain device accountability records documenting the receipt, expiration date, and final disposition (e.g., subject ID if implanted, attempted, or returned to SJM) of all investigational devices. The unique device identifiers and date received must be documented on the log for all valves and delivery systems upon receipt and include the initials of the person completing the log. All devices that are opened must be accounted for on the device accountability log, even if they are not used.

SJM must also maintain device accountability documenting all shipments and returns of investigational devices by unique device identifier, date, and person completing the log. Storage locations for the investigational devices will be locked with access restricted only to investigators or designee.

### 13.18 Economic and Quality of Life Analysis



### 13.19 Publications

Upon receiving Investigational Device Exemption from FDA, the PORTICO clinical study will be registered on <a href="www.clinicaltrials.gov">www.clinicaltrials.gov</a>. The trial will adhere to the publication principles of the International Committee of Medical Journal Editors (ICMJE).



### 13.20 Investigational Site Start-up

### 13.20.1 Study Initiation Visit

Prior to beginning the study, SJM personnel will contact the Investigator to discuss the CIP and review the data requirements in detail.

# 13.20.2 Site Activation 14 Sponsor Contact Information

# 15 Bibliography









# **16 APPENDICES**

# **Appendix A: Abbreviations**

| Abbreviation | Term |
|---|---|
| 6MWT | Six Minute Walk Test |
| AA | Alternative Access |
| ACC | American College of Cardiology |
| ACT | Activated Clotting Time |
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| AF | Atrial Fibrillation |
| AHA | American Heart Association |
| ARB | Angiotensin Receptor Blocker |
| AS | Aortic Stenosis |
| AV | Aortic Valve |
| AVA | Aortic Valve Area |
| AVR | Aortic Valve Replacement |
| BARC | Bleeding Academic Research Consortium |
| BNP | B-type Natriuretic Peptide |
| CAD | Coronary Artery Disease |
| CAP | Continued Access Protocol |
| CAV | FDA Approved and Commercially Available Transcatheter Valve |
| CBC | Complete Blood Count |
| CCS | Canadian Cardiovascular Society |
| CE | Conformité Européene (European Conformity) |
| CEC | Clinical Events Committee |
| CIP | Clinical Investigation Plan |
| CMS | Centers for Medicare & Medicaid Services |
| СРВ | Cardiopulmonary Bypass |
| eCRF | Electronic Case Report Form |
| СТ | Computed Tomography |
| CV | Curriculum Vitae |
| CVA | Cerebral Vascular Accident |
| DSMB | Data Safety Monitoring Board |
| ECG | Electrocardiogram |
| Echo | Echocardiography |
| eDC | Electronic Data Capture |
| EEA | European Economic Area |
| EF | Ejection Fraction |

| Abbreviation | Term |
|---|---|
| EOA | Effective Orifice Area |
| EU | European Union |
| FDA | Food and Drug Administration |
| GI | Gastro Intestinal |
| HOCM | Hypertrophic cardiomyopathy with or without obstruction |
| ICF | Informed Consent Form |
| IDE | Investigational Device Exemption |
| IFU | Instructions For Use |
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| ITT | Intent To Treat |
| KCCQ | Kansas City Cardiomyopathy Questionnaire |
| Kg | Kilogram |
| LBBB | Left Bundle Branch Block |
| LV | Left Ventricular |
| LVEF | Left Ventricular Ejection Fraction |
| MAC | Mitral Annular Calcification |
| MI | Myocardial Infarction |
| MMSE | Mini-mental state examination Mitral Regurgitation Magnetic Resonance Imaging Modified Rankin Scale |
| MR | |
| MRI | |
| mRS | |
| MSCT | Multi-Slice Computed Tomography |
| NCD | National Coverage Determination |
| NIHSS | NIH Stroke Scale |
| NYHA | New York Heart Association |
| PA | Pulmonary Artery |
| PCI | Percutaneous Coronary Intervention |
| PCWP | Pulmonary Capillary Wedge Pressure |
| PI | Principal Investigator |
| QoL | Quality of Life |
| PAVR | Percutaneous Aortic Valve Replacement |
| PMA | Premarket Approval |
| PVD | Peripheral Vascular Disease |
| PVL | Paravalvular Leak |
| RA | Right Atrium |
| RV | Right Ventricular |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |

| Abbreviation | Term |
|--------------|----------------------------------------------|
| SAV | Surgical Aortic Valve |
| SAVR | Surgical Aortic Valve Replacement |
| SD | Standard Deviation |
| SJM | St. Jude Medical, Cardiovascular Division |
| SSC | Subject Selection Committee |
| STS | Society of Thoracic Surgeons |
| TA | Trans Apical |
| TAV | Transcatheter Aortic Valve |
| TAVI | Transcatheter Aortic Valve Implantation |
| TAVR | Transcatheter Aortic Valve Replacement |
| TEE | Transesophageal Echocardiogram (same as TOE) |
| TF | Trans Femoral |
| TIA | Transient Ischemia Attack |
| TAo | Transaortic |
| TTE | Transthoracic Echocardiogram |
| UADE | Unanticipated Adverse Device Effect |
| US | United States (same as USA) |
| USA | United States of America (same as US) |
| VARC 2 | Valve Academic Research Consortium 2 |
| VIV | Valve in Valve |
| WBC | White Blood Cell |
| WMA | World Medical Association |







# **Appendix C: Definitions**

| Source | Definition |
|---|---|
| Cardiovascular | Any one of the following criteria: |
| Mortality | Death due to proximate cardiac cause (e.g. myocardial infarction, cardiac |
| (VARC 2) | tamponade, worsening heart failure) |
| ( | Death caused by non-coronary vascular conditions such as neurological events, |
| | pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other |
| | vascular disease |
| | All procedure-related deaths, including those related to a complication of the |
| | procedure or treatment for a complication of the procedure |
| | All valve-related deaths including structural or nonstructural valve dysfunction or |
| | other valve-related adverse events |
| | Sudden or unwitnessed death |
| | Death of unknown cause |
| Museaudial | |
| Myocardial | Peri-procedural MI (less than or equal to (≤) 72 h after the index procedure) |
| Infarction | New ischemic symptoms (e.g., chest pain or shortness of breath), or new ischemic signs |
| (VARC 2) | (e.g. ventricular arrhythmias, new or worsening heart failure, new ST-segment changes, hemodynamic instability, or imaging evidence of new loss of viable myocardium or new |
| | wall motion abnormality), |
| | AND |
| | Elevated cardiac biomarkers within 72 h after the index procedure consisting of at least |
| | one sample post-procedure with a peak value exceeding 15x upper reference limit |
| | (troponin) or 5x for CK-MB. If cardiac biomarkers are increased at baseline (>99 <sup>th</sup> |
| | percentile), a further increase of at least 50% post-procedure is required AND the peak |
| | value must exceed the previously stated limit. |
| | Spontaneous MI (greater than (>) 72 h after the index procedure) |
| | Any one of the following criteria: |
| | Detection of rise and/or fall of cardiac biomarkers (preferably troponin) with at least |
| | one value above the 99th percentile URL, together with evidence of myocardial |
| | ischemia with at least one of the following: |
| | <ul> <li>Symptoms of ischaemia</li> </ul> |
| | ○ ECG changes indicative of new ischemia [new ST-T changes or new Left Bundle |
| | Branch Block (LBBB)] |
| | <ul> <li>New pathological Q waves in at least two contiguous leads</li> </ul> |
| | <ul> <li>Imaging evidence of new loss of viable myocardium or new wall motion</li> </ul> |
| | abnormality |
| | Sudden, unexpected cardiac death, involving cardiac arrest, often with symptoms |
| | suggestive of myocardial ischemia, and accompanied by presumably new ST-segment |
| | elevation, or new LBBB, and/or evidence of fresh thrombus by coronary angiography |
| | and/ or at autopsy, but death occurring before blood samples could be obtained, or at |
| | a time before the appearance of cardiac biomarkers in the blood. |
| | Pathological findings of an acute myocardial infarction. |
| Stroke | This study is following the FDA's definition of Stroke per FDA's Current Thinking |
| (FDA/VARC 2) | Regarding Neurological Assessments for Transcatheter Valve Trials (Revised: 25 Aug |
| | 2011) and VARC 2 (2012) |
| | 1. Definitions: |
| | a. <u>Stroke</u> : Stroke is an acute episode of focal or global neurological dysfunction caused |
| | by the brain, spinal cord, or retinal vascular injury as a result of hemorrhage or |
| | infarction. |

| Source | Definition |
|---|---|
| - Source | Subclassifications of stroke: |
| | i. <u>Ischemic Stroke</u> is defined as an acute symptomatic episode of focal cerebral, |
| | spinal, or retinal dysfunction caused by an infarction of central nervous system tissue. |
| | ii. <u>Hemorrhagic Stroke</u> is defined as an acute symptomatic episode of focal or global cerebral or spinal dysfunction caused by a nontraumatic |
| | intraparenchymal, intraventricular, or subarachnoid hemorrhage. |
| | Stroke Disability (consistent with VARC 2 Definitions): |
| | i. Disabling: an mRS score of 2 or more at 90 days and an increase of at least one mRS category from an individual's pre-stroke baseline |
| | ii. Non-disabling: an mRS score of < 2 at 90 days or one that does not result in an increase of at least one mRS category from an individual's pre-stroke baseline |
| | b. <u>Cerebral Infarction:</u> Evidence of brain cell death from imaging studies or pathological examination. If there are clinical symptoms, then it is a stroke; otherwise, it is an asymptomatic cerebral infarction. |
| | <ul> <li>c. <u>Transient Ischemic Attack (TIA):</u> A transient (less than (&lt;) 24 hrs) episode of neurological dysfunction caused by focal brain, spinal cord, or retinal ischemia, without acute infarction. No evidence of infarction if imaging performed.</li> <li>d. <u>Encephalopathy:</u> Altered mental state (e.g., seizures, delirium, confusion, hallucinations, dementia, coma, psychiatric episode, etc.).</li> </ul> |
| | e. Intracranial Hemorrhage: Collection of blood between the brain and skull. |
| | Subcategorized as epidural, subdural, and subarachnoid bleeds. |
| Bleeding | Life-threatening or disabling bleeding |
| (VARC 2) | • Fatal bleeding (BARC type 5) <b>OR</b> |
| | <ul> <li>Bleeding in a critical organ, such as intracranial, intraspinal, intraocular, or pericardial<br/>necessitating pericardiocentesis, or intramuscular with compartment syndrome (BARC<br/>type 3b and 3c) OR</li> </ul> |
| | Bleeding causing hypovolemic shock or severe hypotension requiring vasopressors or surgery (BARC type 3b) <b>OR</b> |
| | <ul> <li>Overt source of bleeding with drop in hemoglobin of greater than or equal to (≥) 5 g/dl or whole blood or packed red blood cells (RBCs) transfusion greater than or equal to (≥) 4 U (BARC type 3b). Given 1 U of packed RBC typically will raise blood hemoglobin concentration by 1 g/dl, an estimated decrease in hemoglobin will be calculated.</li> </ul> |
| | Major bleeding (BARC type 3a) |
| | <ul> <li>Overt bleeding either associated with a drop in the hemoglobin level of at least 3.0 g/dl<br/>or requiring transfusion of two or three units of whole blood/ RBC, or causing<br/>hospitalization or permanent injury, or requiring surgery AND</li> </ul> |
| | Does not meet criteria of life-threatening or disabling bleeding |
| | Minor bleeding (BARC type 2 or 3a, depending on the severity) |
| | • Any bleeding worthy of clinical mention (e.g., access site hematoma) that does not |
| | qualify as life-threatening, disabling or major |
| Acute Kidney | Change in serum creatinine (up to 48 h) compared with baseline |
| Injury (AKIN<br>Classification)<br>(VARC 2) | Stage 1 |

| Course | Definition |
|---|---|
| Source | Definition |
| | Increase in serum creatinine to 150% to 199% (1.5 to 1.99 X increase compared with |
| | baseline) or increase of greater than or equal to (≥) 0.3 mg/dl (≥26.4 mmol/l) or |
| | Urine output <0.5 ml/kg per hour for > 6 but < 12 hours |
| | Chang D |
| | Stage 2 |
| | Increase in serum creatinine to 200% to 299% (2.0 to 2.99 X increase compared with |
| | baseline) or |
| | Urine output <0.5 ml/kg per hour for > 12 but < 24 hours |
| | Stage 3 |
| | Increase in serum creatinine to greater than or equal to (≥) 300% (>)3 X increase |
| | compared with baseline) or serum creatinine of $\geq 4.0 \text{ mg/dl}$ ( $\geq 354 \text{ mmol/l}$ ) with an acute |
| | increase of at least 0.5 mg/dl (44 mmol/l) or Urine output < 0.3 ml/kg per hour for ≥ 24 |
| | hours or anuria for ≥ 12 hours. Patients receiving renal replacement therapy are |
| Vacculer | considered to meet Stage 3 criteria irrespective of other criteria. |
| Vascular | Major vascular complications |
| Access Site | Any aortic dissection, aortic rupture, annulus rupture, left ventricle perforation, or |
| and Access-<br>Related | new apical aneurysm/pseudo-aneurysm or |
| Complications | Access site or access-related vascular injury (dissection, stenosis, perforation, |
| (VARC 2) | rupture, arterio-venous fistula, pseudoaneurysm, hematoma, irreversible nerve |
| (VARC 2) | injury, compartment syndrome, percutaneous closure device failure) <i>leading to</i> |
| | death, life-threatening or major bleeding*, visceral ischaemia or neurological |
| | impairment or |
| | Distal embolization (non-cerebral) from a vascular source requiring surgery or |
| | resulting in amputation or irreversible end-organ damage or |
| | The use of unplanned endovascular or surgical intervention associated with death, |
| | major bleeding, visceral ischaemia or neurological impairment or |
| | Any new ipsilateral lower extremity ischemia documented by patient symptoms, |
| | physical exam, and/or decreased or absent blood flow on lower extremity angiogram |
| | or |
| | Surgery for access site-related nerve injury or |
| | Permanent access site-related nerve injury Minor vescular complications |
| | Minor vascular complications |
| | Access site or access-related vascular injury (dissection, stenosis, perforation, |
| | rupture, arterio-venous fistula, pseudoaneuysms, hematomas, percutaneous closure |
| | device failure) <b>not leading to</b> death, life-threatening or major bleeding*, visceral |
| | ischaemia or neurological impairment or |
| | Distal embolization treated with embolectomy and/or thrombectomy and not |
| | resulting in amputation or irreversible end-organ damage or |
| | Any unplanned endovascular stenting or unplanned surgical intervention not |
| | meeting the criteria for a major vascular complication or |
| | Vascular repair or the need for vascular repair (via surgery, ultrasound-guided) |
| | compression, transcatheter embolization, or stent-graft) or |
| | Percutaneous closure device failure |
| | Failure of a closure device to achieve haemostasis at the arteriotomy site leading to |
| | alternative treatment (other than manual compression or adjunctive endovascular |
| | ballooning) |

| Source | Definition | | | |
|---|---|---|---|---|
| Source | Definition - | | | |
| Acute Device<br>Success<br>(VARC 2 with<br>modifications) | <ol> <li>Acute device success defined as: <ul> <li>Absence of procedural mortality</li> <li>Correct positioning of a single prosthetic heart valve into the proper anatomical location</li> <li>Intended performance of the prosthetic heart valve (mean aortic valve gradient &lt;20 mmHg or peak velocity &lt;3 m/s, no moderate or severe prosthetic valve regurgitation)</li> <li>Successful access was obtained as intended by group assignment</li> </ul> </li> <li>Device success is a 'technical' composite endpoint meant to characterize the acute device and procedural factors which underlie vascular access, delivery, and performance of the TAVI system. Echocardiography should be routinely utilized as the standard for measuring prosthetic valve stenosis and regurgitation immediately after TAVI, and should always be performed in a resting state, either within 24–48 h after the index procedure or before hospital discharge.</li> </ol> | | | |
| FDA | Individual Patient Success 1. Acute device success 2. Discharged alive from the hospital without device-related major AEs (Includes AI ≤ 1+) 3. Survival to one year with: O No disabling stroke O No device-or procedure-related mortality O NYHA class ≤ 2, or improvement in NYHA class by at least 1 level from baseline O No re-hospitalizations for valve related complications/dysfunction or CHF due to aortic valve related causes | | | 1 level from |
| Prosthetic<br>Valve Stenosis | conduction abnormal Parameter | | Mild Stenosis | Moderate/<br>severe |
| Criteria In conditions of normal or near normal | Peak velocity (m/s) Mean gradient (mm Hg) | less than (<) 3 | 3–4 | Stenosis greater than (>) 4 greater than |
| stroke volume<br>(50–70 ml).<br>(VARC 2) | Doppler velocity index Effective orifice area | greater than or equal<br>to (≥) 0.35<br>greater than (>) 1.1* | 0.35-0.25 | (>) 40 less than (<) 0.25 less than (<) |
| | (cm²) | | | 0.80 |
| Prosthetic<br>Valve | Diastolic flow reversal in | the descending aorta (sen | ni-quantitative parame | ters) |
| Regurgitation<br>Criteria<br>(VARC 2) | Diastolic flow<br>reversal in the<br>descending aorta<br>PW Doppler | Absent or brief early<br>diastolic | Intermediate | Prominent,<br>holodiastolic |

<sup>\*</sup> Effective orifice area (EOA) used in this protocol is 1.0 cm² for Portico valve of 23mm diameter.

| Source | Definition | | | |
|---|---|---|---|---|
| | Circumferential<br>extent of<br>paraprosthetic AR | less than (<) 10% | 10–29% | greater than or equal ( <u>&gt;</u> ) 30% |
| | Doppler parameters (qua | ntitative) | | |
| | Regurgitant volume<br>(ml/beat) | less than (<) 30% | 30–59% | greater than or equal ( <u>&gt;</u> ) 60% |
| | Regurgitant fraction | less than (<) 30% | 30–49% | greater than or equal ( <u>&gt;</u> ) 50% |
| | EROA (cm²) | 0.10 cm <sup>2</sup> | 0.10-0.29 cm <sup>2</sup> | ≥0.30 cm <sup>2</sup> |

# **Appendix D: Surgical Risk Assessment Tools**

This clinical study requires the use of two surgical risk assessment tools:

- 1. The Society of Thoracic Surgeons' (STS) risk calculation tools, Version 2.73 (<a href="http://riskcalc.sts.org/STSWebRiskCalc273/de.aspx">http://riskcalc.sts.org/STSWebRiskCalc273/de.aspx</a>)
- 2. Euro SCORE II (http://euroscore.org/calc.html)

# Appendix E: Quality of Life - EQ-5D 3L

By placing a checkmark in one box in each group below, please indicate which statements best describe your own health state today.

| Mobility |
|---|
| I have no problems in walking about |
| I have some problems in walking about |
| I am confined to bed |
| Self-Care |
| I have no problems with self-care |
| I have some problems washing or dressing myself |
| I am unable to wash or dress myself |
| <b>Usual Activities</b> (e.g. work, study, housework, family or leisure activities) |
| I have no problems with performing my usual activities |
| I have some problems with performing my usual activities |
| I am unable to perform my usual activities |
| Pain/Discomfort |
| I have no pain or discomfort |
| I have moderate pain or discomfort |
| I have extreme pain or discomfort |
| Anxiety/Depression |
| I am not anxious or depressed |
| I am moderately anxious or depressed |
| I am extremely anxious or depressed |

To help people say how good or bad a health state is, we have drawn a scale (rather like a thermometer) on which the best state you can imagine is marked 100 and the worst state you can imagine is marked 0.



# Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. Thank you for completing this survey!

For each of the following questions, please mark an  $\boxtimes$  in the one box that best describes your answer.

1. In general, would you say your health is:



2. Compared to one year ago, how would you rate your health in general now?

| Much better<br>now than one<br>year ago | Somewhat<br>better<br>now than one<br>year ago | About the same as one year ago | Somewhat<br>worse<br>now than one<br>year ago | Much worse<br>now than one<br>year ago |
|---|---|---|---|---|
| lacktriangle | lacktriangle | lacktriangle | lacktriangle | lacktriangle |
| 1 | 2 | 3 | 4 | 5 |

SF-36v2<sup>®</sup> Health Survey ⊗ 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved.
SF-36° is a registered trademark of Medical Outcomes Trust.
(SF-36v2® Health Survey Standard, United States (English))

| 3. | The following questions are about activities you might do during a typical |
|---|---|
| | day. Does your health now limit you in these activities? If so, how much? |

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not<br>limited<br>at all |
|---|---|---|---|---|
| | Vigorous activities, such as running, lifting heavy objects, participating in strenuous sports | | 2 | 3 |
| ь | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | 1 | 2 | ] з |
| c | Lifting or carrying groceries | 1 | 2 | 3 |
| d | Climbing several flights of stairs | 🗆 1 | 2 | ] з |
| e | Climbing one flight of stairs | 🔲 1 | 2 | ] з |
| f | Bending, kneeling, or stooping | 🗆 1 | 2 | ] з |
| 8 | Walking more than a mile | 🔲 1 | 2 | ] з |
| h | Walking several hundred yards | 🗆 1 | 2 | ] з |
| i | Walking one hundred yards | 🗌 1 | 2 | 3 |
| | Bathing or dressing yourself | Π. | $\Box$ | Π, |

SF-36v2® Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (SF-36v2® Health Survey Standard, United States (English))

| 4. | During the <u>past 4 weeks</u> , how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of your physical health</u> ? | | | | | |
|---|---|---|---|---|---|---|
| | | All of the time | Most of the time | Some of the time | A little of the time | None of<br>the time |
| | Cut down on the <u>amount of</u> <u>time</u> you spent on work or other activities | | 2 | 3 | 4 | 5 |
| ь | Accomplished less than you would like | | 2 | 3 | 4 | 5 |
| e | Were limited in the <u>kind</u> of work or other activities | 1 | 2 | 3 | 4 | 5 |
| d | Had <u>difficulty</u> performing the<br>work or other activities (for<br>example, it took extra effort) | | 2 | 3 | 4 | 5 |
| 5. | During the <u>past 4 weeks</u> ,<br>following problems with y<br>result of any emotional p | your work | or other re | gular daily | activities <u>a</u> | as a |
| | | All of<br>the time | Most of<br>the time | | A little of<br>the time | None of<br>the time |
| | Cut down on the <u>amount of</u><br>time you spent on work or<br>other activities | | 2 | 3 | 4 | s |
| ь | Accomplished less than you would like | 1 | 2 | 3 | 4 | s |
| e | Did work or other activities less carefully than usual | 1 | 2 | 3 | 4 | 5 |

SF-36v2 $^{\rm n}$  Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36 $^{\rm n}$  is a registered trademark of Medical Outcomes Trust. (SF-36v2 $^{\rm n}$  Health Survey Standard, United States (English))

| 6. | During the <u>past 4 weeks</u> , to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? | | | | | | |
|---|---|---|---|---|---|---|---|
| | | Not at all | Slightly | Moderate | ly Qu | ite a bit | Extremely |
| | | <b>V</b> □ 1 | _ 2 | 3 | | <u> </u> | <b>▼</b> |
| 7. | How | v much <u>bo</u> o | <u>dily</u> pain have | you had du | ıring the | e <u>past 4 v</u> | veeks? |
| | | None | Very mild | Mild M | loderate | Severe | Very severe |
| | | <b>▼</b> | 2 | 3 | <b>V</b> □ 4 | 5 | 6 |
| 8. | . During the <u>past 4 weeks</u> , how much did <u>pain</u> interfere with your norm work (including both work outside the home and housework)? | | | | | | |
| | | Not at all | A little bit | Moderate | ly Qu | nite a bit | Extremely |
| | | <b>▼</b> | 2 | 3 | | 4 | <b>▼</b> |

SF-36v2® Health Survey  $\otimes$  1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (SF-36v2® Health Survey Standard, United States (English))
9. These questions are about how you feel and how things have been with you during the past 4 weeks. For each question, please give the one answer that comes closest to the way you have been feeling. How much of the time during the past 4 weeks...

| | All of<br>the time | Most of<br>the time | Some of the time | A little of the time | None of<br>the time |
|---|---|---|---|---|---|
| Did you feel full of life? | | 2 | 3 | | s |
| ь Have you been very nervous? | | 2 | 3 | 4 | 5 |
| Have you felt so down in the<br>dumps that nothing could<br>cheer you up? | | 2 | 3 | 4 | 5 |
| Have you felt calm and peaceful? | 1 | 2 | 3 | 4 | 5 |
| Did you have a lot of energy? | | 2 | 3 | 4 | s |
| Have you felt downhearted and depressed? | 1 | 2 | 3 | 4 | 5 |
| 8 Did you feel worn out? | | 2 | 3 | 4 | 5 |
| h Have you been happy? | | 2 | 3 | 4 | s |
| Did you feel tired? | | 2 | 3 | 4 | 5 |
| 10. During the <u>past 4 weeks</u> ,<br><u>emotional problems</u> inter<br>friends, relatives, etc.)? | | | | | |
| All of Most of the time the time | _ | | A little of<br>the time | None of<br>the time | |
| ▼ ▼ | • | <b>7</b> | $\blacksquare$ | ▼ | |

SF-36v2<sup>®</sup> Health Survey ⊗ 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved.
SF-36° is a registered trademark of Medical Outcomes Trust.
(SF-36v2<sup>®</sup> Health Survey Standard, United States (English))

### 11. How TRUE or FALSE is each of the following statements for you?

| | | Definitely<br>true | Mostly<br>true | Don't<br>know | Mostly<br>false | Definitely<br>false |
|---|---|---|---|---|---|---|
| | | lacksquare | lacksquare | lacksquare | lacksquare | lacksquare |
| * | I seem to get sick a little easier than other people | 🗆 1 | 2 | 3 | 4 | 5 |
| ь | I am as healthy as<br>anybody I know | 🔲 1 | 2 | 3 | 4 | 5 |
| c | I expect my health to get worse | 🗆 1 | 2 | 3 | 4 | 5 |
| d | My health is excellent | 🗌 1 | 2 | 3 | 4 | 5 |

Thank you for completing these questions!

#### Appendix G: Quality of Life – Kansas City Cardiomyopathy Questionnaire (KCCQ)

#### The KC Cardiomyopathy Questionnaire

The following questions refer to your heart failure and how it may affect your life. Please read and complete the following questions. There are no right or wrong answers. Please mark the answer that best applies to you.

Heart failure affects different people in different ways. Some feel shortness of breath while
others feel fatigue. Please indicate how much you are limited by heart failure (shortness of
breath or fatigue) in your ability to do the following activities over the past 2 weeks.

#### Place an X in one box on each line

| Activity | Extremely<br>Limited | Quite a bit<br>Limited | Moderately<br>Limited | Not at all<br>Limited | Limited for<br>other reasons or<br>did not do the<br>activity |
|---|---|---|---|---|---|
| Dressing yourself | | | | | |
| Showering/Bathing | | | | | |
| Walking 1 block on<br>level ground | | | | | |
| Doing yardwork,<br>housework or<br>carrying groceries | | | | | 0 |
| Climbing a flight of<br>stairs without<br>stopping | | | | | |
| Hurrying or jogging (as if to catch a bus) | | | | | |
| Compared with 2 weeks ago, have your symptoms of heart failure (shortness of breath, fatigue, or ankle swelling) changed? My symptoms of heart failure have become Much Slightly Not changed Slightly Much I've had no symptoms worse worse better better over the last 2 weeks | | | | | |

Copyright @1992 -2005 John Spertus, MD, MPH

Original US English

| <ol> <li>Over the past 2<br/>when you woke up</li> </ol> | | times did you have | swelling in y | our feet, ankles ( | or legs |
|---|---|---|---|---|---|
| Every morning | 3 or more times<br>a week, but not<br>every day | 1-2 times a week | Less than o<br>week | | |
| | | | | | 1 |
| 4. Over the past 2 It has been Extremely bothersome | | Moderately bothersome | Slightly bothersome | Not at all bothersome | you?<br>I've had no<br>swelling |
| ш | ь | ш | ы | | |
| 5. Over the past 2<br>what you was | | e, how many times h | as fatigue lii | mited your ability | to do |
| | er day once a day | 3 or more times<br>per week but not<br>every day | per week | Less than once<br>a week | Never over<br>the past 2<br>weeks |
| 6. Over the past 2 | 2 weeks, how much | h has your <b>fatigue</b> b | othered you? | | |
| Extremely bothersome | Quite a bit bothersome | | Slightly<br>othersome | Not at all<br>bothersome | I've had<br>no fatigue<br>□ |
| | weeks, on average<br>hat you wanted? | e, how many times h | as s <b>hortne</b> ss | of breath limite | d your |
| All of the Seve<br>time times pe | | 3 or more times<br>per week but not<br>every day | 1-2 times<br>per week | Less than once<br>a week | Never over<br>the past 2<br>weeks |
| Copyright ⊗1992 –2005 Je | ohn Spertus, MD, MPH | | | Original | US English |

| <ol><li>Over the past</li></ol> | 2 weeks, how n | nuch has your s | hortness of | breath bother | ed you? |
|---|---|---|---|---|---|
| It has been | | | | | |
| Extremely bothersome | Quite a bit bothersome | Moderately<br>bothersome | Slightl<br>botherso | • | |
| in a chair or with | | s to prop you | | | |
| Every night | week, but not ev | | week | a week | past 2 weeks |
| | re symptoms can<br>o do, or whom to | | | | re are you that you |
| Not at all sure | Not very su | re Somewh | _ | Mostly sure | Completely sure |
| 11. How well do | | | | | ur heart failure<br>a low salt diet etc.) |
| Do not understa<br>at all | nd Do not und<br>very w | | omewhat<br>derstand | Mostly<br>understand | Completely<br>understand |
| 12. Over the pas | st 2 weeks, how | nuch has your | heart failur | e limited your | enjoyment of life? |
| It has extremel<br>limited my<br>enjoyment of lif | enjoyment o | f life mod | has<br>erately<br>ted my<br>ent of life | It has slightly<br>limited my<br>enjoyment of li | my enjoyment of |
| | | ,, | | | |
| 13. If you had to spend the rest of your life with your heart failure the way it is <u>right now</u> , how would you feel about this? | | | | | |
| | at all Mo | | newhat | | Completely |
| | sfied dissat | _ | tisfied | satisfied | satisfied |
| Constitute (1902) 2005 | John Courses MC No. | | | | Octobro IVV Tradich |
| Copyright @1992 -2005 | Joint Sperrus, MD, MP1 | 1 | | | Original US English |

| <ol> <li>Over the <u>past</u><br/>your heart fa</li> </ol> | | w often have y | ou felt discou | raged or down in | the dumps t | ecause of |
|---|---|---|---|---|---|---|
| I felt that w<br>all of the ti | ray I felt the<br>me most of | | t that way | I rarely felt that<br>way | I never felt<br>way | that |
| 15. How much does your heart failure affect your lifestyle? Please indicate how your heart failure may have limited your participation in the following activities over the past 2 weeks. | | | | | | |
| | Pleas | se place an X | in one box | on each line | | _ |
| Activity | Severely<br>limited | Limited<br>quite a bit | Moderately<br>limited | Slightly<br>limited | Did not<br>limit at all | Does not<br>apply or did<br>not do for<br>other reasons |
| Hobbies,<br>recreational<br>activities | | | | | | |
| Working or<br>doing household<br>chores | | | | | | |
| Visiting family<br>or friends out of<br>your home | | | | | | |
| Intimate<br>relationships<br>with loved ones | | | | | | |

## Appendix H: Mini-Mental State Examination (MMSE-2)

| MMSI | ~ | Date of examin | ation | | Examiner | | | |
|---|---|---|---|---|---|---|---|---|
| | | Name | | | | Age | Sex | - /1 |
| Standard Vers | ion | Years of school | completed | Purpose of | exam | | | |
| Blue Form | А | ssessment of l | evel of consciousr | ness | | | | |
| | - R | Alert/<br>esponsive | Drowsy | Stuporous | Comatose/<br>Unresponsive | | | |
| in parentheses. A | Administration s<br>o if the response | should be con<br>e is incorrect of | ducted privately | and in the exanuse is correct. Be | to the examinee. It<br>ninee's primary lang<br>gin by introducing<br>your memory. | uage. Unles | | |
| | | | | RE | SPONSE | | SCC | |
| MILK [pause], SE<br>[Repeat up to 3 tire | I am going to | e], BEFORE [ | pause]. Now re | | stop. Ready? Hei<br>ds back to me. | e they are | | e one) |
| | SENSIBLE | | - | | | | 0 | 1 |
| | BEFORE | | - | | | | 0 | 1 |
| | | l. I am going | to ask you to s | av them again | in a few minutes. | | U | |
| ORIENTATION | | | and the second | , | | | | |
| What day is toda | | | | | | | | |
| | vear? | | | | | | 0 | 1 |
| | season? | | | | | | 0 | 1 |
| | month of the y | rear | 4 I I | | | | 0 | 1 |
| | day of the | are Control | <u> </u> | | | | 0 | 1 |
| | date? | | | | | | 0 | 1 |
| ORIENTATION | TO PLACE | te . | | | | | | |
| Where are we no | | | | | | | | |
| | state (or provin | | _ | | | | 0 | 1 |
| | county (or city/ | town)? | _ | | | | 0 | 1 |
| | city/town (or pa | art of city/neig | ghborhood)? | | | | 0 | 1 |
| 1 | building (name | or type)? | | | | | 0 | 1 |
| | floor of the bu | - | _ | | | | 0 | 1 |
| | (room number of<br>ords that are appro | | tting and increasing | gly precise may be | substituted and noted. | | | |
| RECALL | | | · · | , , | | | | |
| What were those | three words I | asked you to | romombor2 [C | o not offer any | hinto 1 | | | |
| | | askeu you it | remember r [L | o not oner any i | riirits.] | | 62753 | |
| | MILK | | ) <del> </del> | | | | 0 | 1 |
| | SENSIBLE<br>BEFORE | | | | | | 0 | 1 |
| | BEFORE | | - | | | | 0 | 1 |
| | If administer<br>the space pro | ing the MMSE<br>ovided at the to | 2-2:SV, copy the Mop of page 2 and c | MMSE-2:BV total total total total adminute with a minute with a minute w | | MSE-2:BV<br>raw score | | |
| PAR • 16204 N | | A CONTRACTOR OF THE PARTY OF TH | | T. 1. 2. | | | 16 max, | |
| MMSE copyright © 1975, 1<br>any form or by any means w<br>9 8 7 6 5 | 998, 2001 and MMSE-<br>rithout written permission | 2 copyright © 2010 to<br>n of PAR. This form is | s printed in blue and burg | jundy ink on white paper | d 2001, 2010 by PAR. May no<br>Any other version is unautho | rized. | | |
| 10/05 | TOCOPYING OR | | Reorder #R | J-6685 | | | Printed i | in the U.S |


| | | MMSE-2:<br>total raw sco | | |
|---|---|---|---|---|
| ATTENTION AND CALCULA | ATION [Serial 7s] | | (16 max | points) |
| Now I'd like you to subtract 7 fr | om 100. Then keep s | subtracting 7 from each answer until I tell you to | o stop. | |
| What is 100 take away 7? | [93] | | 0 | 1 |
| If needed, say: Keep going. | [86] | | 0 | 1 |
| If needed, say: Keep going. | [79] | | 0 | 1 |
| If needed, say: Keep going. | [72] | | 0 | 1 |
| If needed, say: Keep going. | [65] | | 0 | 1 |
| Score 1 point for each correct answe<br>even if the previous answer was inco | | ered correct if it is 7 less than the previous answer, | | |
| NAMING | | | | |
| What is this? [Point to eye.] | | | 0 | 1 |
| What is this? [Point to ear.] | | | 0 | 1 |
| REPETITION | | | | |
| | | dy? IT IS A LOVELY, SUNNY DAY BUT TOO W. ecord response verbatim. Repeat up to one time.] | ARM. | |
| IT IS A LOVELY, SUNNY DAY | BUT TOO WARM. | | 0 | 1 |
| upper half of the detached page, v<br>Use the bottom half of the page as | which has three shapes<br>s a stimulus form for t<br>age as a stimulus and | ge in half along the horizontal perforation line. Use son it, as a stimulus form for the Comprehension the Reading ("CLOSE YOUR EYES") task. Use the response form for the Drawing (intersecting pentagonse form for the Writing take. | ask. | |
| COMPREHENSION | | | | |
| Listen carefully because i am go<br>figures stimulus page.] Look 111<br>and then point to the triangle. | | osc nething. Thou gran new the geometric pint to the irc that point to the quare, | | |
| | Correct response | Observed response | | |
| | 0 | | 0 | 1 |
| | | | 0 | 1 |
| | | | 0 | 1 |
| READING | | | U | |
| Show examinee the word stimulu | s nage 1 Please do v | what this save to do | | |
| CLOSE YOUR | | mat tine says to do. | 0 | 2 |
| CLUSE YOUR I | I I E O | | 0 | 1 |

or spelling.

WRITING

**DRAWING**[Display the intersecting pentagons on the stimulus form and provide a pen or pencil.] Please copy this design. Score 1 point if the drawing consists of two 5-sided figures that intersect to form a 4-sided figure.

[Place the blank piece of paper in front of the examinee and provide a pen or pencil.]

Please write a sentence. [If examinee does not respond, say: Write about where you live.]

Score 1 point if the sentence is comprehensible and contains a subject and a verb. Ignore errors in grammar

| MMSE-2:SV |
|-----------------|
| total raw score |

0

0

30 max, points)

2 WARNING! PHOTOCOPYING OR DUPLICATION OF THIS FORM WITHOUT PERMISSION IS A VIOLATION OF COPYRIGHT LAWS.

# Sample

# **CLOSE YOUR EYES**



# Sample

#### Appendix I: Canadian Cardiovascular Society grading of angina pectoris

Grade I Ordinary physical activity does not cause angina, such as walking and

climbing stairs. Angina with strenuous or rapid or prolonged exertion

at work or recreation

**Grade II** Slight limitation of ordinary activity. Walking or climbing stairs rapidly,

walking uphill, walking or stair climbing after meals, or in cold, or in wind, or under emotional stress, or only during the few hours after awakening. Walking more than two blocks on the level and climbing more than one flight of ordinary stairs at a normal pace and in normal

conditions

Grade III Marked limitation of ordinary physical activity. Walking one or two

blocks on the level and climbing one flight of stairs in normal

conditions and at normal pace

**Grade IV** Inability to carry on any physical activity without discomfort, anginal

syndrome may be present at rest

#### **Appendix J: Frailty Assessment**

The Frailty Index Data Collection Form will be used as an assessment tool to determine if frailty is a high risk factor for subjects prior to enrollment. This assessment will be performed after the informed consent has been obtained and prior to procedure. The assessment can be administered by either an investigator or research coordinator. The frailty assessment consists of three evaluations:

- 1. Katz Index of Independence in Activities of Daily Living
- 2. Grip Strength
- 3. 15 Foot walk test

#### Katz Index of Independence in Activities of Daily Living Activities

| Points (1 or 0) | Independence<br>(1 Point)<br>NO supervision, direction or personal<br>assistance | Dependence<br>(0 Points)<br>WITH supervision, direction,<br>personal assistance or total care |
|---|---|---|
| BATHING Points: | (1 POINT) Bathes self completely or needs<br>help in bathing only a single part of the<br>body such as the back, genital area or<br>disabled extremity | (0 POINTS) Need help with bathing more than one part of the body, getting in or out of the tub or shower. Requires total bathing |
| DRESSING<br>Points: | (1 POINT) Get clothes from closets and drawers and puts on clothes and outer garments complete with fasteners. May have help tying shoes. | (0 POINTS) Needs help with dressing self or needs to be completely dressed. |
| TOILETING Points: | (1 POINT) Goes to toilet, gets on and off, arranges clothes, cleans genital area without help. | (0 POINTS) Needs help transferring to the toilet, cleaning self or uses bedpan or commode. |
| TRANSFERRING Points: | (1 POINT) Moves in and out of bed or chair unassisted. Mechanical transfer aids are acceptable. | (0 POINTS)Needs help in moving from bed to chair or requires a complete transfer. |
| CONTINENCE Points: | (1 POINT) Exercises complete self control over urination and defecation. | (0 POINTS) Is partially or totally incontinent of bowel or bladder. |
| FEEDING<br>Points: | (1 POINT) Gets food from plate into mouth without help. Preparation of food may be done by another person. | (0 POINTS) Needs partial or total help with feeding or requires parenteral feeding. |
| TOTAL Points: | | |

**Grip strength** Subjects elbow should be at a 90 degree angle without arm supported or resting on table or against chest wall. Each grasp should be completed with the dynamometer in the dominant hand.

| Grasp 1 | Grasp 2 | Grasp3 |
|---------|---------|--------|
| Average | | |

# 15 Foot Walk \_\_\_\_\_seconds

| Men | Cutoff for grip strength (Kg) criterion for frailty |
|---|---|
| BMI ≤ 24<br>BMI 24.1-26<br>BMI 26.1-28<br>BMI > 28 | ≤ 29<br>≤ 30<br>≤ 30<br>≤ 32 |
| Women | Cutoff for grip strength (Kg) criterion for frailty |
| BMI ≤ 23<br>BMI 23.1-26<br>BMI 26.1-29<br>BMI > 29 | ≤ 17<br>≤ 17.3<br>≤ 18<br>≤ 21 |
| (Appendix, Fried et al) | |

#### Appendix K: Structured Interview for the Modified Rankin Scale (mRS)

After the NIHSS has been completed, the mRS (by a certified rater) is to be determined and graded by the same certified rater.

The determination of the scale should be made from 5 to 0, i.e., the order presented.

The purpose of the mRS is to record whether the patient is dead, severely, moderately, or slightly disabled and if not dead or disabled, whether the patient is performing all usual activities without symptoms or not. Because subjects and family members may understate the severity of disability, it is important for the rating clinician to understand that the mRS is a clinical scale and not a patient-reported outcome. The rater may ask questions but must assess the disability whether or not in agreement with the subject or family.

"Improving the assessment of outcomes in stroke: use of a structured interview to assign grades on the Modified Rankin Scale" *Stroke*; 33:2243-2246)

5: Severe disability; someone needs to be available at all times; care may be provided by either a trained or an untrained caregiver.

Question: Does the person require constant care?

4: Moderately severe disability; need for assistance with some basic activities of daily living (ADL), but not requiring constant care.

Question: Is assistance essential for eating, using the toilet, daily hygiene, or walking?

3: Moderate disability; need for assistance with some instrumental ADL but not basic ADL.

Question: Is assistance essential for preparing a simple meal, doing household chores, looking after money, shopping, or traveling locally?

2: Slight disability; limitations in participation in usual social roles, but independent for ADL.

Questions: Has there been a change in the person's ability to work or look after others if these were roles before stroke? Has there been a change in the person's ability to participate in previous social and leisure activities? Has the person had problems with relationships or become isolated?

1 No significant disability; symptoms present but not other limitations.

Question: Does the person have difficulty reading or writing, difficulty speaking or finding the right word, problems with balance or coordination, visual problems, numbness (face, arms, legs, hands, feet), loss of movement (face, arms, legs, hands, feet), difficulty with swallowing, or other symptom resulting from stroke?

0 No symptoms at all; no limitations and no symptoms.





#### **Appendix N: NYHA Classification**

Class I Patient has cardiac disease but without resulting limitations of

ordinary physical activity. Ordinary physical activity (e.g., walking several blocks or climbing stairs) does not cause undue fatigue, palpitation, dyspnea, or anginal pain. Limiting symptoms may occur

with marked exertion.

Class II Patient has cardiac disease resulting in slight limitation of ordinary

physical activity. Patient is comfortable at rest. Ordinary physical activity such as walking more than two blocks or climbing more than one flight of stairs results in limiting symptoms (e.g., fatigue,

palpitation, dyspnea, or anginal pain).

Class III Patient has cardiac disease resulting in marked limitation of physical

activity. Patient is comfortable at rest. Less than ordinary physical activity (e.g., walking one to two level blocks or climbing one flight of

stairs) causes fatigue, palpitation, dyspnea, or anginal pain.

**Class IV** Patient has dyspnea at rest that increases with any physical activity.

Patient has cardiac disease resulting in inability to perform any physical activity without discomfort. Symptoms may be present even at rest. If any physical activity is undertaken, discomfort is increased.

#### Appendix O: ATS Guidelines for the Six Minute Walk Test

This Six Minute Walk (6MWT) Test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing.

#### SAFETY ISSUES

- 1. Testing should be performed in a location where a rapid, appropriate response to an emergency is possible. The appropriate location of a crash cart should be determined by the physician supervising the facility.
- 2. Supplies that must be available include oxygen, sublingual nitroglycerine, aspirin, and albuterol (metered dose inhaler or nebulizer). A telephone or other means should be in place to enable a call for help.
- 3. The technician should be certified in cardiopulmonary resuscitation with a minimum of Basic Life Support by an American Health Association—approved cardiopulmonary resuscitation course. Advanced cardiac life support certification is desirable. Training, experience, and certification in related health care fields (registered nurse, registered respiratory therapist, certified pulmonary function technician, etc.) are also desirable. A certified individual should be readily available to respond if needed.
- 4. Physicians are not required to be present during all tests. The physician ordering the test or a supervising laboratory physician may decide whether physician attendance at a specific test is required.
- 5. If a patient is on chronic oxygen therapy, oxygen should be given at their standard rate or as directed by a physician or a protocol.

Reasons for immediately stopping a 6MWT include the following: (1) chest pain, (2) intolerable dyspnea, (3) leg cramps, (4) staggering, (5) diaphoresis, and (6) pale or ashen appearance.

Technicians must be trained to recognize these problems and the appropriate responses. If a test is stopped for any of these reasons, the patient should sit or lie supine as appropriate depending on the severity or the event and the technician's assessment of the severity of the event and the risk of syncope. The following should be obtained based on the judgment of the technician: blood pressure, pulse rate, oxygen saturation, and a physician evaluation. Oxygen should be administered as appropriate.

#### CONTRAINDICATIONS

Absolute contraindications for the 6MWT include the following: unstable angina during the previous month and myocardial infarction during the previous month. Relative contraindications include a resting heart rate of more than 120, a systolic blood pressure of more than 180 mm Hg, and a diastolic blood pressure of more than 100 mm Hg.

Patients with any of these findings should be referred to the physician ordering or supervising the test for individual clinical assessment and a decision about the conduct of the test. The results from a resting electrocardiogram done during the previous 6 months should also be reviewed before testing. Stable exertional angina is not an absolute contraindication for a 6MWT, but patients with these symptoms should perform the test after using their antiangina medication, and rescue nitrate medication should be readily available. A deviation from the Clinical Investigation Plan will need to be collected if the subject is unable to complete this test.

#### LOCATION

The 6MWT should be performed indoors, along a long, flat, straight, enclosed corridor with a hard surface that is seldom traveled. If the weather is comfortable, the test may be performed outdoors. The walking course must be 30 m in length. A 100-ft hallway is, therefore, required. The length of the corridor should be marked every 3 m. The turnaround points should be marked with a cone (such as an orange traffic cone). A starting line, which marks the beginning and end of each 60-m lap, should be marked on the floor using brightly colored tape.

#### **PROCEDURE**

#### REQUIRED EQUIPMENT

- Countdown timer (or stopwatch)
- Mechanical lap counter
- Two small cones to mark the turnaround points
- A chair that can be easily moved along the walking course
- Worksheets on a clipboard
- A source of oxygen
- Sphygmomanometer
- Telephone
- Automated electronic defibrillator

#### PATIENT PREPARATION

- Comfortable clothing should be worn.
- Appropriate shoes for walking should be worn.
- Patients should use their usual walking aids during the test (cane, walker, etc.).
- The patient's usual medical regimen should be continued.
- A light meal is acceptable before early morning or early afternoon tests.
- Patients should not have exercised vigorously within 2 hours of beginning the test.

- This test should be performed about the same time of day for each interval to minimize intraday variability.
- A "warm-up" period before the test should not be performed.
- The patient should sit at rest in a chair, located near the starting position, for at least 10 minutes before the test starts. During this time, check for contraindications, measure pulse and blood pressure, and make sure that clothing and shoes are appropriate. Complete the first portion of the worksheet.

#### **Baseline Measurements**

 Set the lap counter to zero and the timer to 6 minutes. Assemble all necessary equipment (lap counter, timer, clipboard, Borg Scale, worksheet) and move to the starting point.

Instruct the patient as follows:

"The object of this test is to walk as far as possible for 6 minutes. You will walk back and forth in this hallway. Six minutes is a long time to walk, so you will be exerting yourself. You will probably get out of breath or become exhausted. You are permitted to slow down, to stop, and to rest as necessary. You may lean against the wall while resting, but resume walking as soon as you are able.

You will be walking back and forth around the cones. You should pivot briskly around the cones and continue back the other way without hesitation. Now I'm going to show you. Please watch the way I turn without hesitation."

Demonstrate by walking one lap yourself. Walk and pivot around a cone briskly.

"Are you ready to do that? I am going to use this counter to keep track of the number of laps you complete. I will click it each time you turn around at this starting line. Remember that the object is to walk AS FAR AS POSSIBLE for 6 minutes, but don't run or jog.

Start now, or whenever you are ready."

Position the patient at the starting line. You should also stand near the starting line during the test. Do not walk with the patient. As soon as the patient starts to walk, start the timer.

Do not talk to anyone during the walk. Use an even tone of voice when using the standard phrases of encouragement. Watch the patient. Do not get distracted and lose count of the laps. Each time the participant returns to the starting line, click the lap counter once (or mark the lap on the worksheet). Let the participant see you do it. Exaggerate the click using body language, like using a stopwatch at a race.

After the first minute, tell the patient the following (in even tones):

"You are doing well. You have 5 minutes to go."

When the timer shows 4 minutes remaining, tell the patient the following: "Keep up the good work. You have 4 minutes to go."

When the timer shows 3 minutes remaining, tell the patient the following:

"You are doing well. You are halfway done."

When the timer shows 2 minutes remaining, tell the patient the following: "Keep up the good work. You have only 2 minutes left."

When the timer shows only 1 minute remaining, tell the patient:

"You are doing well. You have only 1 minute to go."

Do not use other words of encouragement (or body language to speed up).

If the patient stops walking during the test and needs a rest, say this:

"You can lean against the wall if you would like; then continue walking whenever you feel able."

Do not stop the timer. If the patient stops before the 6 minutes are up and refuses to continue (or you decide that they should not continue), wheel the chair over for the patient to sit on, discontinue the walk, and note on the worksheet the distance, the time stopped, and the reason for stopping prematurely.

When the timer is 15 seconds from completion, say this:

"In a moment I'm going to tell you to stop. When I do, just stop right where you are and I will come to you."

When the timer rings (or buzzes), say this: "Stop!"

Walk over to the patient. Consider taking the chair if they look exhausted. Mark the spot where they stopped.

## Appendix P: Barthel Index

| THE | Patient Name: | | |
|---|---|---|---|
| BARTHEL | Rater Name: | | |
| INDEX | Date: | | |
| Activity | | | Score |
| FEEDING 0 = unable 5 = needs help cutting, spreading butt 10 = independent | er, etc., or requires modified diet | | |
| BATHING<br>0 = dependent<br>5 = independent (or in shower) | | | |
| GROOMING 0 = needs to help with personal care 5 = independent face/hair/teeth/shavir | ng (implements provided) | | |
| DRESSING 0 = dependent 5 = needs help but can do about half u 10 = independent (including buttons, | | | |
| BOWELS 0 = incontinent (or needs to be given of 5 = occasional accident 10 = continent | enemas) | | |
| BLADDER 0 = incontinent, or catheterized and up 5 = occasional accident 10 = continent | nable to manage alone | | |
| TOILET USE 0 = dependent 5 = needs some help, but can do some 10 = independent (on and off, dressin | | | |
| TRANSFERS (BED TO CHAIR AND II 0 = unable, no sitting balance 5 = major help (one or two people, ph 10 = minor help (verbal or physical) 15 = independent | | | |
| MOBILITY (ON LEVEL SURFACES) 0 = immobile or < 50 yards 5 = wheelchair independent, including 10 = walks with help of one person (v 15 = independent (but may use any ai | g corners, > 50 yards<br>erbal or physical) > 50 yards | | |
| STAIRS | a, 101 e. manipio, ononje oo jaras | | |
| 0 = unable<br>5 = needs help (verbal, physical, carry<br>10 = independent | ring aid) | | |
| | | TOTAL (0-100): | 1 <u>2</u> |

 ${\it Provided by the Internet Stroke Center-www.strokecenter.org}$ 

#### The Barthel ADL Index: Guidelines

- 1. The index should be used as a record of what a patient does, not as a record of what a patient could do.
- The main aim is to establish degree of independence from any help, physical or verbal, however minor and for whatever reason.
- 3. The need for supervision renders the patient not independent.
- 4. A patient's performance should be established using the best available evidence. Asking the patient, friends/relatives and nurses are the usual sources, but direct observation and common sense are also important. However direct testing is not needed.
- Usually the patient's performance over the preceding 24-48 hours is important, but occasionally longer periods will be relevant.
- 6. Middle categories imply that the patient supplies over 50 per cent of the effort.
- 7. Use of aids to be independent is allowed.

#### References

Mahoney FI, Barthel D. "Functional evaluation: the Barthel Index." Maryland State Medical Journal 1965;14:56-61. Used with permission.

Loewen SC, Anderson BA. "Predictors of stroke outcome using objective measurement scales." *Stroke.* 1990;21:78-81.

Gresham GE, Phillips TF, Labi ML. "ADL status in stroke: relative merits of three standard indexes." Arch Phys Med Rehabil. 1980;61:355-358.

Collin C, Wade DT, Davies S, Horne V. "The Barthel ADL Index: a reliability study." *Int Disability Study*. 1988;10:61-63.

#### **Copyright Information**

The Maryland State Medical Society holds the copyright for the Barthel Index. It may be used freely for non-commercial purposes with the following citation:

Mahoney FI, Barthel D. "Functional evaluation: the Barthel Index." Maryland State Med Journal 1965;14:56-61. Used with permission.

Permission is required to modify the Barthel Index or to use it for commercial purposes.

Provided by the Internet Stroke Center — www.strokecenter.org









































































## Appendix U: NIH Stroke Scale (NIHSS)



| Patient id | lentification | | | _ |
|------------|-------------------|-----|-----|---|
| | Pt. Date of Birth | _/_ | _/_ | _ |
| Hospital _ | | | | |
| | Date of Exam | | | |

| <u> </u> | Hospital ( | _ |
|---|---|---|
| SCALE | Date of Exam/_ | |
| Interval: [] Baseline [] 2 hours post treatment [] 24 ho | | |
| Time:: []am []pm | | |
| Person Administering Scale | | |
| Administer stroke scale items in the order listed. Record plack and change scores. Follow directions provided for earth what the clinician thinks the patient can do. The clinician sl | ch exam technique. Scores should reflect what the patier | nt does, no |
| Except where indicated, the patient should not be coached ( | i.e., repeated requests to patient to make a special effort). | |
| Instructions | Scale Definition | Score |
| Level of Consciousness: The investigator must choose a response if a full evaluation is prevented by such obstacles as an endotracheal tube, language barrier, orotracheal trauma/bandages. A 3 is scored only if the patient makes no movement (other than reflexive). | | |

1b. LOC Questions: The patient is asked the month and his/her age. The answer must be correct - there is no partial credit for being close. Aphasic and stuporous patients who do not comprehend the questions will score 2. Patients unable to speak because of endotracheal intubation, orotracheal trauma, severe dysarthria from any cause, language barrier, or any other problem not secondary to aphasia are given a 1. It is important that only the initial answer be graded and that the examiner not "help" the patient with verbal or non-verbal cues.

posturing) in response to noxious stimulation.

Answers both questions correctly.

make movements (not stereotyped). 3 - Responds only with reflex motor or autonomic effects or totally unresponsive, flaccid, and areflexic.

obtunded and requires strong or painful stimulation to

- 1 Answers one question correctly.
- 2 Answers neither question correctly.
- 1c. LOC Commands: The patient is asked to open and close the eyes and then to grip and release the non-paretic hand. Substitute another one step command if the hands cannot be used. Credit is given if an unequivocal attempt is made but not completed due to weakness. If the patient does not respond to command, the task should be demonstrated to him or her (pantomime), and the result scored (i.e., follows none, one or two commands). Patients with trauma, amputation, or other physical impediments should be given sultable one-step commands. Only the first attempt is scored.
- 0 Performs both tasks correctly.
- 1 Performs one task correctly.
- 2 Performs neither task correctly.
- 2. Best Gaze: Only horizontal eye movements will be tested. Voluntary or reflexive (oculocephalic) eye movements will be scored, but caloric testing is not done. If the patient has a conjugate deviation of the eyes that can be overcome by voluntary or reflexive activity, the score will be 1. If a patient has an isolated peripheral nerve paresis (CN III, IV or VI), score a 1. Gaze is testable in all aphasic patients. Patients with ocular trauma, bandages, pre-existing blindness, or other disorder of visual aculty or fields should be tested with reflexive movements, and a choice made by the investigator. Establishing eye contact and then moving about the patient from side to side will occasionally clarify the presence of a partial gaze palsy.
- 0 Normal.
- 1 Partial gaze palsy; gaze is abnormal in one or both eyes, but forced deviation or total gaze paresis is not present.
- 2 Forced deviation, or total gaze paresis not overcome by the oculocephalic maneuver.



| NIH | Patient Identification | |
|---|---|---|
| STROKE | Pt. Date of Birth/ | |
| | Hospital( | ) |
| SCALE | Date of Exam/ | _/ |
| [] 3 months [] Other | ours post onset of symptoms ±20 minutes [] 7-10 days () 0 - No visual loss. | |
| confrontation, using finger counting or visual threat, as appropriate.<br>Patients may be encouraged, but if they look at the side of the<br>moving fingers appropriately, this can be scored as normal. If there is<br>unliateral blindness or enucleation, visual fields in the remaining eye<br>are scored. Score 1 only if a clear-cut asymmetry, including<br>quadrantanopia, is found. If patient is blind from any cause, score 3.<br>Double simultaneous stimulation is performed at this point. If there is<br>extinction, patient receives a 1, and the results are used to respond to<br>Item 11. | Partial hemianopia. Complete hemianopia. Bilateral hemianopia (blind including cortical blindness). | |
| 4. Facial Palsy: Ask – or use pantomime to encourage – the patient to show teeth or raise eyebrows and close eyes. Score symmetry of grimace in response to noxious stimuli in the poorly responsive or non-comprehending patient. If facial trauma/bandages, orotracheal tube, tape or other physical barriers obscure the face, these should be removed to the extent possible. | Normal symmetrical movements. Minor paralysis (flattened nasolablal fold, asymmetry on smilling). Partial paralysis (total or near-total paralysis of lower face). Complete paralysis of one or both sides (absence of facial movement in the upper and lower face). | _ |
| 5. Motor Arm: The limb is placed in the appropriate position: extend the arms (paims down) 90 degrees (if sitting) or 45 degrees (if supine). Drift is scored if the arm falls before 10 seconds. The aphasic patient is encouraged using urgency in the voice and pantomime, but not noxious stimulation. Each limb is tested in turn, beginning with the non-paretic arm. Only in the case of amputation or joint fusion at the shoulder, the examiner should record the score as untestable (UN), and clearly write the explanation for this choice. | No drift; limb holds 90 (or 45) degrees for full 10 seconds. Drift; limb holds 90 (or 45) degrees, but drifts down before full 10 seconds; does not hit bed or other support. Some effort against gravity; limb cannot get to or maintain (if cued) 90 (or 45) degrees, drifts down to bed, but has some effort against gravity. No effort against gravity; limb falls. No movement. UN – Amputation or joint fusion, explain: Sa. Left Arm Sb. Right Arm | |
| 6. Motor Leg: The limb is placed in the appropriate position: hold the leg at 30 degrees (always tested supine). Drift is scored if the leg falls before 5 seconds. The aphasic patient is encouraged using urgency in the voice and pantomime, but not noxious stimulation. Each limb is tested in turn, beginning with the non-paretic leg. Only in the case of amputation or joint fusion at the hip, the examiner should record the score as untestable (UN), and clearly write the explanation for this choice. | No drift; leg holds 30-degree position for full 5 seconds. Drift; leg falls by the end of the 5-second period but does not hit bed. Some effort against gravity; leg falls to bed by 5 seconds, but has some effort against gravity. No effort against gravity; leg falls to bed immediately. No movement. UN = Amputation or joint fusion, explain: | |



| Patient | Identification | | | _ |
|----------|---------------------|---|---|---|
| | Pt. Date of Birth _ | | 1 | |
| Hospital | | ( | | |
| | Date of Exam _ | | | _ |

| | Hospital( | |
|---|---|---|
| SCALE | Date of Exam/ | _/ |
| Interval: [] Baseline [] 2 hours post treatment [] 24 ho<br>[] 3 months [] Other | ours post onset of symptoms ±20 minutes [] 7-10 days | _ |
| 7. Limb Ataxia: This item is aimed at finding evidence of a unilateral cerebellar lesion. Test with eyes open. In case of visual defect, ensure testing is done in intact visual field. The finger-nose-finger and heel-shin tests are performed on both sides, and ataxia is scored only if present out of proportion to weakness. Ataxia is absent in the patient who cannot understand or is paralyzed. Only in the case of amputation or joint fusion, the examiner should record the score as untestable (UN), and clearly write the explanation for this choice. In case of bilindness, test by having the patient touch nose from extended arm position. | 0 - Absent. 1 - Present in one limb. 2 - Present in two limbs. UN - Amputation or joint fusion, explain: | |
| 8. Sensory: Sensation or grimace to pinprick when tested, or withdrawal from noxious stimulus in the obtunded or aphasic patient. Only sensory loss attributed to stroke is scored as abnormal and the examiner should test as many body areas (arms [not hands], legs, trunk, face) as needed to accurately check for hemisensory loss. A score of 2, "severe or total sensory loss," should only be given when a severe or total loss of sensation can be clearly demonstrated. Stuporous and aphasic patients will, therefore, probably score 1 or 0. The patient with brainstem stroke who has bilateral loss of sensation is scored 2. If the patient does not respond and is quadriplegic, score 2. Patients in a coma (Item 1a-3) are automatically given a 2 on this Item. | Normal; no sensory loss; patient feels pinprick is less sharp or is dull on the affected side; or there is a loss of superficial pain with pinprick, but patient is aware of being touched. Severe to total sensory loss; patient is not aware of being touched in the face, arm, and leg. | |
| 9. Best Language: A great deal of information about comprehension will be obtained during the preceding sections of the examination. For this scale item, the patient is asked to describe what is happening in the attached picture, to name the items on the attached naming sheet and to read from the attached list of sentences. Comprehension is judged from responses here, as well as to all of the commands in the preceding general neurological exam. If visual loss interferes with the tests, ask the patient to identify objects placed in the hand, repeat, and produce speech. The intuibated patient should be asked to write. The patient in a coma (item 1a-3) will automatically score 3 on this item. The examiner must choose a score for the patient with stupor or limited cooperation, but a score of 3 should be used only if the patient is mute and follows no one-step commands. | No aphasia; normal. Mild-to-moderate aphasia; some obvious loss of fluency or facility of comprehension, without significant limitation on Ideas expressed or form of expression. Reduction of speech and/or comprehension, however, makes conversation about provided materials difficult or impossible. For example, in conversation about provided materials, examiner can identify picture or naming card content from patient's response. 2 - Severe aphasia; all communication is through fragmentary expression; great need for inference, questioning, and guessing by the listener. Range of information that can be exchanged is limited; listener carries burden of communication. Examiner cannot identify materials provided from patient response. 3 - Mute, global aphasia; no usable speech or auditory comprehension. | |
| 10. Dysarthria: If patient is thought to be normal, an adequate sample of speech must be obtained by asking patient to read or repeat words from the attached list. If the patient has severe aphasia, the clarity of articulation of spontaneous speech can be rated. Only if the patient is intubated or has other physical parriers to producing speech, the examiner should record the score as untestable (UN), and clearly write an explanation for this choice. Do not tell the patient why he or she is being tested. | O = Normal. Mild-to-moderate dysarthria; patient siurs at least some words and, at worst, can be understood with some difficulty. Severe dysarthria; patient's speech is so siurred as to be unintelligible in the absence of or out of proportion to any dysphasia, or is mute/anarthric. UN = Intubated or other physical barrier, explain: | |



| NIH | Patient Identification. | |
|---|---|---|
| STROKE | Pt. Date of Birth/ | _/ |
| SCALE | Hospital( | |
| Interval: [] Baseline [] 2 hours post treatment [] 24 ho<br>[] 3 months [] Other | | |
| 11. Extinction and inattention (formerly Neglect): Sufficient Information to Identify neglect may be obtained during the prior testing. If the patient has a severe visual loss preventing visual double simultaneous stimulation, and the cutaneous stimuli are normal, the score is normal. If the patient has aphasia but does appear to attend to both sides, the score is normal. The presence of visual spatial neglect or anosagnosia may also be taken as evidence of abnormality. Since the abnormality is scored only if present, the item is never untestable. | O - No abnormality. 1 - Visual, tactile, auditory, spatial, or personal inattention or extinction to bilateral simultaneous stimulation in one of the sensory modalities. 2 - Profound hemi-inattention or extinction to more than one modality; does not recognize own hand or orients to only one side of space. | |



You know how.

Down to earth.

I got home from work.

Near the table in the dining room.

They heard him speak on the radio last night.



**MAMA** 

TIP - TOP

FIFTY - FIFTY

**THANKS** 

**HUCKLEBERRY** 

**BASEBALL PLAYER** 





<sup>&</sup>lt;sup>1</sup> Kappetein AP, Head SJ, Genereux P, et al. Updated Standardized Endpoint Definitions for Transcatheter Aortic Valve Implantation: The Valve Academic Research Consortium-2 Consensus Document. J Am Coll Cardiol 2012;60:1438-1454.






# Appendix W: Portico IDE FlexNav Study Synopsis

# 1. PURPOSE

#### 1.1 Indications for Use

The Portico™ valve is indicated for transcatheter delivery in patients with symptomatic severe native aortic stenosis who are considered high or extreme surgical risk.

The FlexNav<sup>™</sup> delivery system is indicated for transcatheter delivery of the Portico<sup>™</sup> valve. The delivery system is indicated for insertion into the vessel with or without an arterial introducer sheath.

The FlexNav<sup>™</sup> loading system is indicated for loading the Portico<sup>™</sup> valve in the FlexNav<sup>™</sup> delivery system.

# 1.2 Study Design and Objectives

The primary objective of the PORTICO pivotal IDE FlexNav study ("FlexNav study") is to characterize the safety of the second-generation FlexNav™ Delivery System ("FlexNav™ Delivery System).

The FlexNav study will be conducted as a prospective, multicenter, investigational study arm of the PORTICO pivotal IDE trial. Up to 200 patients (includes a maximum of 100 roll-ins) with symptomatic, severe aortic stenosis considered by a local Heart Team to be high or extreme risk for surgical aortic valve implantation will be enrolled from up to 70 US and Australian IDE sites. Upon provision of informed consent, subjects will undergo Portico valve implantation via a transfemoral or alternative access approach. Subject selection and key data collection will follow the pivotal IDE protocol to facilitate direct comparison of safety outcomes with the randomized cohort.



# 1.3 Study Endpoints

# 1.3.1 Primary Endpoint

The primary safety endpoint of the FlexNav study is VARC II defined major vascular complications at 30 days.



#### 1.3.2 Descriptive Endpoints

A selection of endpoints from the pivotal IDE trial including valve performance parameters, clinical function assessments and adverse events defined according to VARC II<sup>1</sup> criteria will be assessed at 30 days and included in the PMA application:

# **Descriptive Endpoints:**

- Non-hierarchical composite of all-cause mortality, disabling stroke, life threatening bleeding requiring blood transfusion, acute kidney injury requiring dialysis, or major vascular complications at 30 days from the index procedure
- 2. All-cause mortality at 30 days from the index procedure
- 3. Disabling stroke at 30 days from the index procedure
- 4. Non-disabling stroke at 30 days from the index procedure
- 5. Life threatening bleeding requiring blood transfusion at 30 days from the index procedure
- 6. Major bleeding at 30 days from the index procedure
- 7. Acute kidney injury at 30 days from the index procedure
- 8. Minor vascular complication rates at 30 days from the index procedure
- 9. Permanent pacemaker insertion at 30 days from the index procedure
- 10. Paravalvular Leak (PVL) at 30 days from the index procedure
- 11. NYHA functional classification at 30 days from the index procedure
- 12. KCCQ Quality of Life (QOL) score from baseline to 30 days from the index procedure
- 13. Technical device success defined as successful vascular access, delivery and deployment of the Portico Valve; retrieval with the delivery system and correct positioning of a single valve in the proper anatomical location

Additional endpoints to be assessed at one year but not included in the PMA application:

- Composite of all-cause mortality or disabling stroke at one year from the index procedure
- 2. All-cause mortality at one year from the index procedure
- Disabling stroke at one year from the index procedure
- 4. Non-disabling stroke at one year from the index procedure
- 5. Paravalvular Leak (PVL) at one year from the index procedure
- 6. KCCQ Quality of Life (QOL) score from baseline and one year from the index procedure
- 7. NYHA functional classification at one year from the index procedure

#### 2. CLINICAL PROTOCOL

# 2.1 Background Information

In 2017, the AHA/ACC revised their guidelines in a focused update to make TAVR a class I indication (previously a class IIa indication) for the treatment of aortic valve stenosis in patients at prohibitive or high-surgical risk.<sup>2</sup> As the use of TAVR expands into younger, lower risk populations, minimizing vascular complications which are amongst the most frequent and serious complications of TAVR is of paramount importance as studies show vascular and bleeding complications during the procedure are associated with increased morbidity and mortality risk.<sup>3,4</sup>

Edwards LifeSciences and Medtronic are the current TAVR market leaders accounting for 95% of the global TAVI market share. Two key design elements of the commercially-available balloon-expandable Edwards Sapian 3 valve and self-expanding Medtronic CoreValve Evolut R/Pro valve systems that help mitigate the frequency of vascular and bleeding complications are: 1) a low insertion profile due to the use of a custom expandable sheath (Sapien 3) and integrated sheath (Evolut R/Pro); and 2) the ability to achieve precise valve placement without repositioning or with minimal need to resheath and reposition.

The safety and effectiveness of the Abbott (legacy St. Jude Medical) family of CE Marked Portico™ Transcatheter Aortic Heart Valves (size range 23-29mm) is currently being assessed in the PORTICO pivotal US IDE trial.

The proposed FlexNav study will be conducted as separate arm of the pivotal IDE trial and will include a minimum of 100 analysis patients.

Characterizing the safety profile of the FlexNav<sup>™</sup> Delivery system with respect to rate of major vascular complications, which is expected to be directly impacted by the recent design modifications to the delivery system, is the primary focus of the clinical investigation.

#### 2.2 Rationale

The rationale for conducting the FlexNav study within the PORTICO pivotal IDE trial is to enable the direct comparison of 30-day safety outcomes data for the FlexNav™ Delivery System to the first-generation Portico Delivery System. Results from the FlexNav study will be included in a PMA application to support US approval of the Portico Transcatheter Heart Valve and FlexNav™ Delivery System.





## 3.3 Instructions for Use

For instructions for use (IFU) of the Portico™ Transcatheter Aortic Heart Valve and FlexNav™ Delivery System please refer to the IFU (Number 600014467) which includes the following:

- Portico™ Transcatheter Aortic Valve (PRT-23-IDE, PRT-25-IDE, PRT-27-IDE, PRT-29-IDE)
- FlexNav<sup>TM</sup> Delivery System (FN-DS-SM-IDE, FN-DS-LG-IDE)
- FlexNav<sup>TM</sup> Loading System (FN-LS-SM-IDE, FN-LS-LG-IDE)





#### 4. RISK AND BENEFITS OF THE STUDY DEVICE AND CLINICAL STUDY

There are no changes to the risk or benefits reported in the pivotal IDE trial for subjects participating in the FlexNav Study. Please refer to the Portico™ Transcatheter Aortic Heart Valve and FlexNav Delivery System IFU for a description of risk to benefits and a list of the potential adverse events.

#### 5. STUDY POPULATION

## 5.1 Study Cohort

The FlexNav study is limited to subjects with symptomatic, severe aortic stenosis who are determined to be at high or extreme operative risk for surgical aortic valve replacement. The operative risk determination will be based on the Society of Thoracic Surgeons (STS) Adult Cardiac Surgery Risk Calculator. A surgeon's assessment of operative comorbidities, including medical and anatomic factors not captured by the STS risk calculator will also be considered in determining a subject's operative risk.



#### 5.2 Inclusion/Exclusion Criteria

The inclusion/exclusion criteria for the FlexNav Study is the same as the pivotal IDE trial. Refer to Sections 5.1 and 5.2 of the main protocol for details.

Additional exclusion criteria for subjects being considered for Portico valve implantation via an alternative access approach using the FlexNav™ Delivery System include:

For transaortic access using the FlexNav™ Delivery System:

- 1. Subject has a distance between the annular plane and the aortic access site <7 cm (2.8")
- 2. Subject has a distance between the annular plane and the separate introducer sheath distal tip <6 cm (2.4")

For subclavian/axillary access using the FlexNav™ Delivery System:

- 1. Subject's access vessel (subclavian/axillary) has a distance between the annular plane and the integrated sheath distal tip <17 cm (6.7")
- 2. Subject's access vessel requires the delivery system to be advanced through a separate introduce sheath

## 5.3 Screening Process

Subject case reviews will be conducted to determine a patient's eligibility to receive a Portico valve (roll-in and analysis population) by the same independent Subject Selection Committee used in the pivotal IDE trial.

The risk definitions will be the same as the pivotal IDE trial to ensure a consistent patient population is enrolled. The Subject Selection Committee will provide final determination of a subject's risk classification and primary access approach. If a site disagrees with the Subject Selection Committee's final decision regarding risk classification and/or primary access approach the subject will not be eligible for enrollment in the study.

#### 6. SUBJECT ASSIGNMENTS

Subjects in the FlexNav study are not randomized. All subjects will undergo a Portico valve implant attempt.

Subject assignments (roll-in or analysis population) will be assigned by the Sponsor after Subject Selection Committee approval and prior to enrollment, based on the primary implanting physician's recent Portico experience.

## 6.1 Subject Enrollment

Subjects will be considered enrolled into the FlexNav study after completion of all of the following steps:

- 1. Signed informed consent is obtained.
- 2. Based on the screening assessments, it is determined that the subject meets all of the inclusion and none of the exclusion criteria.
- 3. Subject is approved by the Subject Selection Committee.
- 4. Subject assignment (roll-in or analysis) has been determined by the Sponsor.
- 5. The Portico delivery system enters the subjects' body.

Subjects who are approved by the Subject Selection Committee to receive a Portico valve via transfemoral access and are found during the procedure not to be suitable for this delivery modality (per the heart team medical decision) may receive a Portico valve using an alternate access modality and vice versa. This will be considered a protocol deviation unless the Subject Selection Committee pre-approved the subject for multiple access sites. The rationale for this decision must be documented by the site.



#### 6.2 Roll-in Cohort

A minimum of one (1) and up to three (3) roll-in subjects will be required per primary implanting physician at each site. Data from roll-in subjects will be added to the IDE Roll-in Registry and will not be included in the analysis population of 100 subjects. A maximum of 100 roll-in subjects will be permitted in the study.

The total number of roll-in subjects required per site will be at the discretion of the Sponsor and will be based on the primary implanting physician's recent Portico implant experience.

# 6.3 Proctoring

### 7. STUDY CONDUCT

Assessments required at screening, baseline, pre- and post-procedure, prior to hospital discharge and during follow-up in the FlexNav study will be the same as that in the pivotal IDE trial. Stroke ascertainment and evaluation will be performed according to VARC II recommendations and the pivotal IDE protocol. Detailed information can be found in Section 7.0 of the main protocol.

Subjects enrolled in the FlexNav study will be followed for a minimum of one year and annually thereafter for up to 5 years.

#### 7.1 Core Laboratories

independent core laboratories and processes used in the pivotal IDE trial will be utilized for evaluating CT images, ECG rhythms and echocardiograms for the FlexNav study.

## 7.2 Subject Selection Committee

The independent Subject Selection Committee will be responsible for final approval of a study subjects':

1. risk classification (high vs extreme) based on patients' clinical history, STS score, non-STS comorbidities (including frailty indices) and key patient demographics.

2. primary access route based on independent core-laboratory CT imaging. A secondary access route may also be approved.

As in the pivotal IDE trial, the Subject Selection Committee will provide guidance with respect to Portico valve size selection based on CT-measured annular dimensions (area, perimeter, diameter, eccentricity) and calcification. However, the investigational site has the final decision for which Portico valve size is selected for implantation.

#### 8. DATA COLLECTION AND MANAGEMENT

The schedule for data collection and management of data will follow the pivotal IDE trial. Refer to Section 8.0 of the main protocol for details.

Enrolled subjects who undergo a Portico implant attempt but do not receive a Portico valve will be assessed for any adverse events through to 30 days post-procedure, and will then be terminated from the study.

If a subject is consented and undergoes study-specific testing (i.e., testing that would not be done if they were not being considered for the study) but is not enrolled in the study (FlexNav™ Delivery System does not enter the subject's body), the subject will be exited from the study without any further follow-up.

#### 9. INDEPENDENT BOARDS

#### 9.1 Clinical Events Committee

All adverse events will be adjudicated by the same independent Clinical Events Committee used in the pivotal IDE trial according to the Valve Academic Research Consortium (VARC II) definitions<sup>1</sup>. The independent Clinical Events Committee will have final adjudication responsibilities for subject outcomes related to the primary safety endpoint at 30 days and descriptive endpoints at 30 days and one-year follow-up.

The independent Clinical Events Committee will be responsible for adjudicating the following adverse events at 30 days:

- mortality (all-cause and cardiovascular related)
- stroke (non-disabling and disabling)
- life-threatening bleeding requiring blood transfusion
- major bleeding
- acute kidney injury requiring dialysis
- major vascular complications (access-site related and access related)
- minor vascular complications
- permanent pacemaker insertion

The independent Clinical Events Committee will be responsible for adjudicating the following adverse events at one year:

mortality (all-cause and cardiovascular related)

• stroke (non-disabling and disabling)

# 9.2 Data and Safety Monitoring Board

independent Data and Safety Monitoring Board used in the pivotal IDE trial will be engaged to review the progress and safety of subjects enrolled in the FlexNav study.

# **10. STATISTICAL METHODS AND ANALYSIS**



# 10.3 Primary Endpoint

Acceptable safety of the FlexNav™ Delivery System will be determined from a predefined precision estimate for VARC II-defined major vascular complications at 30 days. Results will be summarized and descriptively compared in context of results for the first-generation Delivery System in the randomized cohort (Portico arm) of the pivotal IDE trial.

A comparison to published results for the Portico valve and latest-generation commercially- available transcatheter valves will also be provided.

# **10.4 Descriptive Endpoints**

Descriptive endpoints will be summarized and presented for the analysis population (n=100 subjects) and according to access route (transfemoral vs alternative access). Additionally, all descriptive endpoints at 30 days will be summarized and descriptively compared to rates reported in the randomized cohort of the pivotal IDE trial as well as published results for Portico and latest-generation commercially available valves.



# 11.0 Bibliography








































